CLINICAL TRIAL: NCT02257567
Title: A Phase IB/II Study Evaluating The Safety, Tolerability and Anti-Tumor Activity of Polatuzumab Vedotin in Combination With Rituximab (R) or Obinutuzumab (G) Plus Bendamustine (B) in Relapsed or Refractory Follicular or Diffuse Large B-Cell Lymphoma
Brief Title: A Study of Polatuzumab Vedotin (DCDS4501A) in Combination With Rituximab or Obinutuzumab Plus Bendamustine in Participants With Relapsed or Refractory Follicular or Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29365; 2014-001361-28 (EudraCT Number)
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Bendamustine Hydrochloride; obinutuzumab; polatuzumab vedotin; Fluid Therapy; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Arm A (Phase II Randomization): Polatuzumab+BR in FL (Experimental): Polatuzumab vedotin will be administered with bendamustine and rituximab in participants with FL.
  Interventions: Drug: Bendamustine; Drug: Polatuzumab vedotin (Liquid); Drug: Rituximab
- Arm B (Phase II Randomization): BR in FL (Active Comparator): Bendamustine and rituximab will be administered alone (that is, without polatuzumab vedotin) as a control arm in participants with FL.
  Interventions: Drug: Bendamustine; Drug: Rituximab
- Arm C (Phase II Randomization): Polatuzumab+BR in DLBCL (Experimental): Polatuzumab vedotin will be administered with bendamustine and rituximab in participants with DLBCL.
  Interventions: Drug: Bendamustine; Drug: Polatuzumab vedotin (Liquid); Drug: Rituximab
- Arm D (Phase II Randomization): BR in DLBCL (Active Comparator): Bendamustine and rituximab will be administered alone (that is, without polatuzumab vedotin) as a control arm in participants with DLBCL.
  Interventions: Drug: Bendamustine; Drug: Rituximab
- Arm E (Phase II Expansion): Polatuzumab+BG in FL (Experimental): Polatuzumab vedotin will be administered with bendamustine and obinutuzumab in participants with FL.
  Interventions: Drug: Bendamustine; Drug: Obinutuzumab; Drug: Polatuzumab vedotin (Liquid)
- Arm F (Phase II Expansion): Polatuzumab+BG in DLBCL (Experimental): Polatuzumab vedotin will be administered with bendamustine and obinutuzumab in participants with DLBCL.
  Interventions: Drug: Bendamustine; Drug: Obinutuzumab; Drug: Polatuzumab vedotin (Liquid)
- Cohort 1A (Phase Ib Safety Run-In): Polatuzumab+BR in DLBCL (Experimental): Polatuzumab vedotin will be administered with bendamustine and rituximab in participants with DLBCL.
  Interventions: Drug: Bendamustine; Drug: Polatuzumab vedotin (Liquid); Drug: Rituximab
- Cohort 1A (Phase Ib Safety Run-In): Polatuzumab+BR in FL (Experimental): Polatuzumab vedotin will be administered with bendamustine and rituximab in participants with FL.
  Interventions: Drug: Bendamustine; Drug: Polatuzumab vedotin (Liquid); Drug: Rituximab
- Cohort 1B (Phase Ib Safety Run-In): Polatuzumab+BG in DLBCL (Experimental): Polatuzumab vedotin will be administered with bendamustine and obinutuzumab in participants with DLBCL.
  Interventions: Drug: Bendamustine; Drug: Obinutuzumab; Drug: Polatuzumab vedotin (Liquid)
- Cohort 1B (Phase Ib Safety Run-In): Polatuzumab+BG in FL (Experimental): Polatuzumab vedotin will be administered with bendamustine and obinutuzumab in participants with FL.
  Interventions: Drug: Bendamustine; Drug: Obinutuzumab; Drug: Polatuzumab vedotin (Liquid)
- Arm G (Phase II NF Cohort): Polatuzumab+BR in DLBCL (Experimental): In this New Formulation (NF) cohort, Polatuzumab vedotin (lyophilized) will be administered with bendamustine and rituximab in participants with DLBCL.
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Polatuzumab vedotin (Lyophilized)
- Arm H (Phase II NF Cohort): Polatuzumab+BR in DLBCL (Experimental): In this NF cohort, Polatuzumab vedotin (lyophilized) will be administered with bendamustine and rituximab in participants with DLBCL.
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Polatuzumab vedotin (Lyophilized)

INTERVENTIONS:
Drug: Bendamustine — Bendamustine 90 milligrams per meter-squared (mg/m^2) per day administered IV on Days 2 and 3 of Cycle 1, then on Days 1 and 2 of each subsequent cycle for up to 6 cycles (each cycle is 21 days in DLBCL and 28 days in FL).
  Other Names: Treanda; Ribomustin; Levact
Drug: Obinutuzumab — Obinutuzumab 1000 milligrams (mg) IV on Days 1, 8, and 15 of Cycle 1 and on Day 1 of each subsequent cycle for up to 6 cycles (each cycle is 21 days in DLBCL and 28 days in FL).
  Other Names: GA101; Gazyva; Gazyvaro
  Arms: Arm E (Phase II Expansion): Polatuzumab+BG in FL; Arm F (Phase II Expansion): Polatuzumab+BG in DLBCL; Cohort 1B (Phase Ib Safety Run-In): Polatuzumab+BG in DLBCL; Cohort 1B (Phase Ib Safety Run-In): Polatuzumab+BG in FL
Drug: Polatuzumab vedotin (Liquid) — Polatuzumab vedotin 1.8 milligrams per kilogram (mg/kg) administered IV on Day 2 of Cycle 1, then on Day 1 of each subsequent cycle for up to 6 cycles (each cycle is 21 days in DLBCL and 28 days in FL).
  Other Names: DCDS4501A
  Arms: Arm A (Phase II Randomization): Polatuzumab+BR in FL; Arm C (Phase II Randomization): Polatuzumab+BR in DLBCL; Arm E (Phase II Expansion): Polatuzumab+BG in FL; Arm F (Phase II Expansion): Polatuzumab+BG in DLBCL; Cohort 1A (Phase Ib Safety Run-In): Polatuzumab+BR in DLBCL; Cohort 1A (Phase Ib Safety Run-In): Polatuzumab+BR in FL; Cohort 1B (Phase Ib Safety Run-In): Polatuzumab+BG in DLBCL; Cohort 1B (Phase Ib Safety Run-In): Polatuzumab+BG in FL
Drug: Rituximab — Rituximab standard dose, 375 mg/m^2 IV on Day 1 of each cycle for up to 6 cycles (each cycle is 21 days in DLBCL and 28 days in FL).
  Other Names: Rituxan; MabThera
  Arms: Arm A (Phase II Randomization): Polatuzumab+BR in FL; Arm B (Phase II Randomization): BR in FL; Arm C (Phase II Randomization): Polatuzumab+BR in DLBCL; Arm D (Phase II Randomization): BR in DLBCL; Arm G (Phase II NF Cohort): Polatuzumab+BR in DLBCL; Arm H (Phase II NF Cohort): Polatuzumab+BR in DLBCL; Cohort 1A (Phase Ib Safety Run-In): Polatuzumab+BR in DLBCL; Cohort 1A (Phase Ib Safety Run-In): Polatuzumab+BR in FL
Drug: Polatuzumab vedotin (Lyophilized) — Participants in the New Formulation (NF) Cohort (Arms G and H) will follow the same schedule and dosing requirements as participants in the other Phase II cohorts (Arms A-F).
  Other Names: DCDS4501S
  Arms: Arm G (Phase II NF Cohort): Polatuzumab+BR in DLBCL; Arm H (Phase II NF Cohort): Polatuzumab+BR in DLBCL

SUMMARY:
This study is a multicenter, open-label study of polatuzumab vedotin administered by intravenous (IV) infusion in combination with standard doses of bendamustine (B) and rituximab (R) or obinutuzumab (G) in participants with relapsed or refractory follicular lymphoma (FL) or diffuse large B-cell lymphoma (DLBCL). The study comprises two stages: a Phase Ib safety run-in stage and a Phase II stage. The anticipated time on treatment is 18 weeks for participants with DLBCL and 24 weeks for participants with FL.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed relapsed or refractory FL (Grades 1, 2, or 3a) or relapsed or refractory DLBCL
* If the participant has received prior bendamustine, response duration must have been greater than (>) 1 year (for participants who have relapse disease after a prior regimen)
* At least one bi-dimensionally measurable lesion on imaging scan defined as >1.5 centimeters (cm) in its longest dimension
* Confirmed availability of archival or freshly collected tumor tissue
* The Phase II NF Cohorts (Arms G and H) will be required to submit tissue and pathology report for central pathology review.
* Life expectancy of at least 24 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Adequate hematological function unless inadequate function is due to underlying disease

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies (MAbs, or recombinant antibody-related fusion proteins) or known sensitivity or allergy to murine products
* Contraindication to bendamustine, rituximab, or obinutuzumab
* Prior use of any MAb, radioimmunoconjugate, or antibody-drug conjugate (ADC) within 4 weeks or 5 half-lives before Cycle 1 Day 1
* Treatment with radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy, or any investigational agent for the purposes of treating cancer within 2 weeks prior to Cycle 1 Day 1
* Ongoing corticosteroid use >30 mg per day prednisone or equivalent, for purposes other than lymphoma symptom control
* Completion of autologous stem cell transplant (SCT) within 100 days prior to Cycle 1 Day 1
* Prior allogeneic SCT
* Eligibility for autologous SCT
* Grade 3b FL
* History of transformation of indolent disease to DLBCL
* Primary or secondary CNS lymphoma
* Current Grade >1 peripheral neuropathy
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina) or significant pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection requiring treatment with IV antibiotics or hospitalization within 4 weeks prior to Cycle 1 Day 1
* Suspected or latent tuberculosis
* Positive test results for chronic hepatitis B virus (HBV) infection or for hepatitis C virus (HCV) antibody
* Known history of human immunodeficiency virus (HIV) seropositive status or known infection with human T-cell leukemia virus 1 (HTLV-1) virus
* Women who are pregnant or lactating or who intend to become pregnant within a year of the last dose of study treatment in the rituximab cohort or within 18 months of last dose in the obinutuzumab cohort
* Evidence of laboratory abnormalities in standard renal, hepatic, or coagulation function tests
* Treatment with chimeric antigen receptor T-cell therapy within 100 days prior to Cycle 1, Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (62):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Univ of Colorado Canc Ctr, Aurora, Colorado
  - Cancer Specialists; North Florida ;Jacksonville (AC Skinner Pkwy), Jacksonville, Florida
  - Emory Univ Winship Cancer Inst, Atlanta, Georgia
  - Joliet Oncology-Hematology; Associates, Ltd., Joliet, Illinois
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - Weinberg CA Inst Franklin Sq, Baltimore, Maryland
  - Regional Cancer Care Associates LLC - Morristown, Morristown, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - West Clinic, Germantown, Tennessee
  - Swedish Cancer Inst., Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Australia (4):
  - Prince of Wales Hospital; Oncology, Randwick, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Monash Medical Centre; Haematology Research, Clayton, Victoria
- Canada (4):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre; Oncology, Halifax, Nova Scotia
  - Hopital Maisonneuve- Rosemont; Oncology, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Czechia (4):
  - Fakultni nemocnice Brno; Interni hematologicka a onkologicka klinika, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultní nemocnice Ostrava Klinika hematoonkologie, Ostrava
  - I Interni klinika; Vseobecna fakultni nemocnice, Prague
- France (6):
  - Chu Site Du Bocage;Hematologie Clinique, Dijon
  - Centre Hospitalier Departemental Les Oudairies, La Roche-sur-Yon
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - CHU Saint Eloi; Service d'Hématologie Clinique, Montpellier
  - CHU Lyon Sud - Service Hématologie, Pierre-Bénite
  - Centre Henri Becquerel; Hematologie, Rouen
- Germany (5):
  - HELIOS Klinikum Erfurt - Innere Medizin - 4. Medizinische Klinik, Hämatologie, Erfurt
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Abt. für Hämatologie und Onkologie, Mainz
  - Joh. Wesling Klinikum Minden; Klinik fuer Hämatologie und Onkologie, Minden
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Klinik der Uni Regensburg; Hämatologie/Onkologie, Studienzentrale, Regensburg
- Hungary (3):
  - Semmelweis University, First Dept of Medicine, Budapest
  - National Institute of Oncology, A Dept of Internal Medicine, Budapest
  - University of Debrecen Medical and Health Science Center, Institute of Internal medicine Building B, Debrecen
- Italy (4):
  - Istituto Nazionale Tumori Irccs Fondazione g. Pascale;s.c. Ematologia Oncologica, Napoli, Campania
  - A.O. Spedali Civili Di Brescia-P.O. Spedali Civili;U.O. Ematologia, Brescia, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Emato-Oncologia, Milan, Lombardy
  - Ospedale Civile SS. Antonio E Biagio DI Alessandria; Ematologia, Alessandria, Piedmont
- UMC St. Radboud; Hematology, Nijmegen, Netherlands
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Hospital Universitari Vall d'Hebron; Servicio de Hematologia, Barcelona
  - Hospital Clinic i Provincial de Barcelona; Hematology, Barcelona
  - Hospital Universitario la Paz; Servicio de Hematologia, Madrid
  - Hospital Clinico Universitario de Salamanca;Servicio de Hematologia, Salamanca
  - Hospital Universitario Virgen del Rocio; Servicio de Hematologia, Seville
- Turkey (Türkiye) (4):
  - Ankara University; Hematology, Ankara
  - Dokuz Eylul Uni ; Hematology, Izmir
  - Ondokuzmayis University Medical Faculty Heamatology Department, Samsun
  - Karadeniz Technical Uni School of Medicine; Hematology, Trabzon
- United Kingdom (4):
  - KINGS COLLEGE HOSPITAL; Commercial R&D Amendments, Kings Health Partners Clinical Trials Office, London
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester
  - Nottingham City Hospital; Dept of Haematology, Nottingham
  - Southampton General Hospital; Somers Cancer Research Building, Southampton

REFERENCES:
- [Derived] Jemaa S, Ounadjela S, Wang X, El-Galaly TC, Kostakoglu L, Knapp A, Ku G, Musick L, Sahin D, Wei MC, Yin S, Bengtsson T, De Crespigny A, Carano RAD. Automated Lugano Metabolic Response Assessment in 18F-Fluorodeoxyglucose-Avid Non-Hodgkin Lymphoma With Deep Learning on 18F-Fluorodeoxyglucose-Positron Emission Tomography. J Clin Oncol. 2024 Sep 1;42(25):2966-2977. doi: 10.1200/JCO.23.01978. Epub 2024 Jun 6. PMID 38843483
- [Derived] Bosch F, Kuruvilla J, Vassilakopoulos TP, Maio DD, Wei MC, Zumofen MB, Nastoupil LJ. Indirect Treatment Comparisons of Mosunetuzumab With Third- and Later-Line Treatments for Relapsed/Refractory Follicular Lymphoma. Clin Lymphoma Myeloma Leuk. 2024 Feb;24(2):105-121. doi: 10.1016/j.clml.2023.09.007. Epub 2023 Sep 28. PMID 37981564
- [Derived] Herrera AF, Tracy S, Croft B, Opat S, Ray J, Lovejoy AF, Musick L, Paulson JN, Sehn LH, Jiang Y. Risk profiling of patients with relapsed/refractory diffuse large B-cell lymphoma by measuring circulating tumor DNA. Blood Adv. 2022 Mar 22;6(6):1651-1660. doi: 10.1182/bloodadvances.2021006415. PMID 35086141
- [Derived] Sehn LH, Hertzberg M, Opat S, Herrera AF, Assouline S, Flowers CR, Kim TM, McMillan A, Ozcan M, Safar V, Salles G, Ku G, Hirata J, Chang YM, Musick L, Matasar MJ. Polatuzumab vedotin plus bendamustine and rituximab in relapsed/refractory DLBCL: survival update and new extension cohort data. Blood Adv. 2022 Jan 25;6(2):533-543. doi: 10.1182/bloodadvances.2021005794. PMID 34749395
- [Derived] Betts KA, Thuresson PO, Felizzi F, Du EX, Dieye I, Li J, Schulz M, Masaquel AS. US cost-effectiveness of polatuzumab vedotin, bendamustine and rituximab in diffuse large B-cell lymphoma. J Comp Eff Res. 2020 Oct;9(14):1003-1015. doi: 10.2217/cer-2020-0057. Epub 2020 Oct 8. PMID 33028076
- [Derived] Shi R, Lu T, Ku G, Ding H, Saito T, Gibiansky L, Agarwal P, Li X, Jin JY, Girish S, Miles D, Li C, Lu D. Asian race and origin have no clinically meaningful effects on polatuzumab vedotin pharmacokinetics in patients with relapsed/refractory B-cell non-Hodgkin lymphoma. Cancer Chemother Pharmacol. 2020 Sep;86(3):347-359. doi: 10.1007/s00280-020-04119-8. Epub 2020 Aug 8. PMID 32770353
- [Derived] Lu T, Gibiansky L, Li X, Li C, Shi R, Agarwal P, Hirata J, Miles D, Chanu P, Girish S, Jin JY, Lu D. Exposure-safety and exposure-efficacy analyses of polatuzumab vedotin in patients with relapsed or refractory diffuse large B-cell lymphoma. Leuk Lymphoma. 2020 Dec;61(12):2905-2914. doi: 10.1080/10428194.2020.1795154. Epub 2020 Jul 24. PMID 32705923
- [Derived] Sehn LH, Herrera AF, Flowers CR, Kamdar MK, McMillan A, Hertzberg M, Assouline S, Kim TM, Kim WS, Ozcan M, Hirata J, Penuel E, Paulson JN, Cheng J, Ku G, Matasar MJ. Polatuzumab Vedotin in Relapsed or Refractory Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2020 Jan 10;38(2):155-165. doi: 10.1200/JCO.19.00172. Epub 2019 Nov 6. PMID 31693429

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 331 participants with relapsed or refractory (R/R) follicular lymphoma (FL) or diffuse large B cell lymphoma (DLBCL) were enrolled in this study at 56 investigative sites in the following countries: Australia, Canada, Czech Republic, France, Germany, Hungary, Italy, Korea, the Netherlands, Spain, Turkey, United Kingdom, and the United States from 15 October 2014 to 21 October 2021.
Pre-assignment Details: Participants were enrolled in Phase Ib and Phase II to receive polatuzumab vedotin (pola) (liquid formulation in randomized & expansion stages; lyophilized formulation in new formulation (NF) cohorts) in combination with standard doses of bendamustine (B) & rituximab (R)/obinutuzumab (G). Out of 331 participants, 327 participants received at least one dose of study drug and their intended treatment.
Groups:
- Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL: Participants with FL received pola, 1.8 milligrams per kilogram (mg/kg), as intravenous (IV) infusion on Day 2 of Cycle 1 (each cycle is 28 days), and thereafter on Day 1 of Cycles 2 to 6. Participants also received bendamustine 90 milligrams per meter-squared (mg/m^2), as IV infusion on Days 2 and 3 of Cycle 1, and thereafter on Days 1 and 2 of Cycles 2 to 6 and rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1 to 6, in combination with pola.
- Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL: Participants with DLBCL received pola, 1.8 mg/kg, as IV infusion on Day 2 of Cycle 1 (each cycle is 21 days), and thereafter on Day 1 of Cycles 2 to 6. Participants also received bendamustine, 90 mg/m^2, as IV infusion on Days 2 and 3 of Cycle 1, and thereafter on Days 1 and 2 of Cycles 2 to 6 and rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1 to 6, in combination with pola.
- Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL; Arm E (Phase II Expansion): Pola+BG in FL: Participants with FL received pola, 1.8 mg/kg, as IV infusion on Day 2 of Cycle 1 (each cycle is 28 days), and thereafter on Day 1 of Cycles 2 to 6. Participants also received bendamustine 90 mg/m^2, as IV infusion on Days 2 and 3 of Cycle 1, and thereafter on Days 1 and 2 of Cycles 2 to 6 and obinutuzumab 1000 mg, as IV infusion on Days 1, 8, and 15 of Cycle 1 and on Day 1 of Cycles 2 to 6 in combination with pola.
- Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL; Arm F (Phase II Expansion): Pola+BG in DLBCL: Participants with DLBCL received pola, 1.8 mg/kg, as IV infusion on Day 2 of Cycle 1 (each cycle is 21 days), and thereafter on Day 1 of Cycles 2 to 6. Participants also received bendamustine 90 mg/m^2, as IV infusion on Days 2 and 3 of Cycle 1, and thereafter on Days 1 and 2 of Cycles 2 to 6 and obinutuzumab 1000 mg, as IV infusion on Days 1, 8, and 15 of Cycle 1 and on Day 1 of Cycles 2 to 6 in combination with pola.
- Arm A (Phase II Randomization): Pola+BR in FL: Participants with FL received pola, 1.8 mg/kg, as IV infusion on Day 2 of Cycle 1 (each cycle is 28 days), and thereafter on Day 1 of Cycles 2 to 6. Participants also received bendamustine 90 mg/m^2, as IV infusion on Days 2 and 3 of Cycle 1, and thereafter on Days 1 and 2 of Cycles 2 to 6 and rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1 to 6, in combination with pola.
- Arm B (Phase II Randomization): BR in FL: Participants with FL received bendamustine 90 mg/m^2, as IV infusion on Days 2 and 3 of Cycle 1 (each cycle is 28 days), thereafter on Days 1 and 2 of Cycles 2 to 6 in combination with rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1 to 6.
- Arm C (Phase II Randomization): Pola+BR in DLBCL: Participants with DLBCL received pola, 1.8 mg/kg, as IV infusion on Day 2 of Cycle 1 (each cycle is 21 days), and thereafter on Day 1 of Cycles 2 to 6. Participants also received bendamustine 90 mg/m^2, as IV infusion on Days 2 and 3 of Cycle 1, and thereafter on Days 1 and 2 of Cycles 2 to 6 and rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1 to 6, in combination with pola.
- Arm D (Phase II Randomization): BR in DLBCL: Participants with DLBCL received bendamustine 90 mg/m^2, as IV infusion on Days 2 and 3 of Cycle 1 (each cycle is 21 days), thereafter on Days 1 and 2 of Cycles 2 to 6 in combination with rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1 to 6.
- Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL: Participants with DLBCL received pola (lyophilized formulation), 1.8 mg/kg, as IV infusion on Day 2 of Cycle 1 (each cycle is 21 days), and thereafter on Day 1 of Cycles 2 to 6. Participants also received bendamustine 90 mg/m^2, as IV infusion on Days 2 and 3 of Cycle 1, and thereafter on Days 1 and 2 of Cycles 2 to 6 and rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1 to 6, in combination with pola.
Period: Overall Study
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Started | 6 | 6 | 6 | 6 | 39 | 41 | 40 | 40 | 20 | 21 | 106
Safety Population (Safety population was defined as all participants who have received at least one dose of study medication.) | 6 | 6 | 6 | 6 | 38 | 41 | 39 | 39 | 20 | 20 | 106
Completed | 4 | 4 | 2 | 1 | 20 | 22 | 6 | 2 | 16 | 0 | 30
Not Completed | 2 | 2 | 4 | 5 | 19 | 19 | 34 | 38 | 4 | 21 | 76
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 2 | 2 | 2 | 4 | 15 | 11 | 26 | 30 | 2 | 18 | 65
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 1
Not completed — Not treated/Per Sponsor Participant Could not Continue/Pathology Showed Transformation: Cycle 1Day 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 6 | 6 | 6 | 1 | 1 | 10

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized, whether or not the participants received the assigned treatment.
Groups:
- Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL; Arm A (Phase II Randomization): Pola+BR in FL: Participants with FL received pola, 1.8 mg/kg, as IV infusion on Day 2 of Cycle 1 (each cycle is 28 days), and thereafter on Day 1 of Cycles 2 to 6. Participants also received bendamustine 90 mg/m^2, as IV infusion on Days 2 and 3 of Cycle 1, and thereafter on Days 1 and 2 of Cycles 2 to 6 and rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1 to 6, in combination with pola.
- Total: Total of all reporting groups
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 39 | 41 | 40 | 40 | 20 | 21 | 106 | 331
Age, Continuous [Median (Full Range); unit: years] | 68.0 [54 to 73] | 65.0 [58 to 79] | 63.5 [42 to 73] | 71.0 [53 to 84] | 65.0 [37 to 74] | 63.0 [39 to 80] | 67.0 [33 to 86] | 71.0 [30 to 84] | 60.5 [37 to 86] | 65.0 [26 to 86] | 70.0 [24 to 94] | 67.0 [24 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 1 | 18 | 23 | 12 | 15 | 10 | 10 | 54 | 151
  Male | 2 | 4 | 4 | 5 | 21 | 18 | 28 | 25 | 10 | 11 | 52 | 180
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 1 | 0 | 0 | 1 | 2 | 6 | 4 | 1 | 6 | 8 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 2 | 0 | 1 | 7
  White | 5 | 5 | 6 | 6 | 33 | 33 | 26 | 31 | 16 | 15 | 83 | 259
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 4 | 6 | 5 | 4 | 1 | 0 | 14 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 3 | 2 | 3 | 14
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 34 | 34 | 35 | 36 | 16 | 19 | 87 | 285
  Not Stated | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 1 | 0 | 0 | 13 | 22
  Unknown | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 1 | 0 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. AEs were reported based on the National Cancer Institute Common Terminology Criteria for AEs, version 4.0 (NCI-CTCAE, v4.0).
Time Frame: From the study start up to the end of the study (up to approximately 84 months)
Population: Safety population consisted of all ITT participants from Phase Ib who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of participants | 100 | 100 | 100 | 100

2. Primary Outcome: Arm G+H (Phase II NF Cohort): Percentage of Participants With AEs
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as AEs. AEs were reported based on the NCI-CTCAE, v4.0. As pre-specified in the protocol data reported is combined for Arms G and H. Values have been rounded off to the nearest whole number.
Time Frame: From Month 37 to Month 84 (up to approximately 47 months)
Population: Safety population consisted of all ITT participants from Arms G+H (Phase II NF Cohort) who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 106
percentage of participants | 99.1

3. Primary Outcome: Cohort 1a (Phase Ib): Percentage of Participants With Treatment Emergent Anti-Drug Antibodies (ADAs) to Polatuzumab Vedotin
Description: The number of participants with positive results for ADA against pola at Baseline and at any of the post-baseline assessment time-points were reported. Participants positive at any post-baseline time points were post-baseline evaluable participants determined to have "Treatment-induced ADAs" or "Treatment-enhanced ADA" during the study period. Treatment-induced ADA = negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at baseline who has one or more post-baseline titer results that are at least 0.60 titer unit (t.u.) greater than the baseline titer result. Treatment emergent ADA is the sum of treatment-induced ADAs and treatment enhanced ADAs. Values have been rounded off to the nearest whole number.
Time Frame: Baseline up to approximately Month 24
Population: Safety population consisted of all ITT participants from Cohort 1a (Phase Ib) who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL
Number analyzed (Participants) | 6 | 6
percentage of participants
  Baseline Prevalence of ADAs | 50.0 | 33.3
  Post-Baseline Incidence of ADAs | 0 | 33.3

4. Primary Outcome: Cohort 1b (Phase Ib): Percentage of Participants With Treatment Emergent ADAs to Polatuzumab Vedotin and Obinutuzumab
Description: The number of participants with positive results for ADA against pola and obinutuzumab at Baseline and at any of the post-baseline assessment time-points were reported. Participants positive at any post-baseline time points were post-baseline evaluable participants determined to have "Treatment-induced ADAs" or "Treatment-enhanced ADA" during the study period. Treatment-induced ADA = negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at baseline who has one or more post-baseline titer results that are at least 0.60 t.u. greater than the baseline titer result. Treatment emergent ADA is the sum of treatment-induced ADAs and treatment enhanced ADAs. Values have been rounded off to the nearest whole number.
Time Frame: Baseline up to approximately Month 24
Population: Safety population consisted of all ITT participants from Cohort 1b (Phase Ib) who received at least one dose of study medication. 'Number Analyzed' is the number of participants with data available for analysis at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL
Number analyzed (Participants) | 6 | 6
percentage of participants
  Baseline Prevalence of ADAs to Polatuzumab vedotin | 0 | 0
  Post-Baseline Incidence of ADAs to Polatuzumab vedotin | 0 | 0
  Baseline Prevalence of ADAs to Obinutuzumab: number analyzed (Participants) | 6 | 5
  Baseline Prevalence of ADAs to Obinutuzumab | 0 | 0
  Post-Baseline Incidence of ADA to Obinutuzumab | 0 | 0

5. Primary Outcome: Arms G+H: (Phase II NF Cohorts): Percentage of Participants With Treatment Emergent ADAs to Polatuzumab Vedotin (Lyophilized)
Description: The number of participants with positive results for ADA against lyophilized pola at Baseline and at any of the post-baseline assessment time-points were reported. Participants positive at any post-baseline time points were post-baseline evaluable participants determined to have "Treatment-induced ADAs" or "Treatment-enhanced ADA" during the study period. Treatment-induced ADA = negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at baseline who has one or more post-baseline titer results that are at least 0.60 t.u. greater than the baseline titer result. Treatment emergent ADA is the sum of treatment-induced ADAs and treatment enhanced ADAs. Values have been rounded off to the nearest whole number.
Time Frame: From Month 37 to Month 84 (up to approximately 47 months)
Population: Safety population consisted of all ITT participants from Arm G+H (Phase II NF cohort) who received at least one dose of study medication. 'Overall Number Analyzed' is the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoint.
Measure: Number; unit: percentage of participants
Groups:
- Arm G (Phase II NF Cohort): Pola+BR in DLBCL; Arm H (Phase II NF Cohort): Pola+BR in DLBCL: Participants with DLBCL received pola (lyophilized formulation), 1.8 mg/kg, as IV infusion on Day 2 of Cycle 1 (each cycle is 21 days), and thereafter on Day 1 of Cycles 2 to 6. Participants also received bendamustine 90 mg/m^2, as IV infusion on Days 2 and 3 of Cycle 1, and thereafter on Days 1 and 2 of Cycles 2 to 6 and rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1 to 6, in combination with pola.
Arm/Group | Arm G (Phase II NF Cohort): Pola+BR in DLBCL | Arm H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 41 | 62
percentage of participants
  Baseline Prevalence of ADAs to Polatuzumab | 0.0 | 1.6
  Post-Baseline Incidence of ADAs to Polatuzumab: number analyzed (Participants) | 39 | 60
  Post-Baseline Incidence of ADAs to Polatuzumab | 2.6 | 5.0

6. Primary Outcome: Phase II Randomized and NF Cohorts: Percentage of Participants With Complete Response (CR) at Primary Response Assessment (PRA) Based on Positron Emission Tomography (PET)-Computed Tomography (CT) Scan as Determined by Independent Review Committee (IRC)
Description: CR was assessed by IRC at PRA according to Modified Lugano Response Criteria (MLRC). Per MLRC, CR based on PET-CT was defined as complete metabolic response (MR) in lymph nodes and extralymphatic sites (ELS) with a score of 1, 2, or 3 with or without residual mass, on 5-point scale (5PS) where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake > mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow. Bone marrow is normal by morphology; if indeterminate, immunohistochemistry (IHC) negative. As pre-specified in the protocol data reported is combined for Arms G and H. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts and 28 days for FL cohorts) or after final dose of study treatment. Values have been rounded off to the nearest whole number.
Time Frame: 6 to 8 weeks after Cycle 6 Day 1 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts) or last dose of study drug (up to approximately 28 weeks)
Population: ITT population included all randomized participants in Phase II Randomized and NF cohorts irrespective of whether or not they received the study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 39 | 41 | 40 | 40 | 106
percentage of participants | 69.2 [52.43 to 82.98] | 63.4 [46.94 to 77.88] | 42.5 [27.04 to 59.11] | 17.5 [7.34 to 32.78] | 39.6 [30.25 to 49.59]
Statistical Analysis 1: Comparison: Arm A (Phase II Randomization): Pola+BR in FL vs Arm B (Phase II Randomization): BR in FL; Test type: Superiority; p = 0.5353, Cochran-Mantel-Haenszel; Difference in Response Rates = 5.82, 95% CI 2-sided [-14.53 to 25.38]
Statistical Analysis 2: Comparison: Arm C (Phase II Randomization): Pola+BR in DLBCL vs Arm D (Phase II Randomization): BR in DLBCL; Test type: Superiority; p = 0.0128, Cochran-Mantel-Haenszel; Difference in Response Rates (4.89 = 25.00, 95% CI 2-sided [4.89 to 42.63]

7. Primary Outcome: Arm H (Phase II NF Cohort): Percentage of Participants With CR at PRA Based on PET-CT as Determined by the IRC
Description: CR was assessed by IRC at PRA according to MLRC. Per MLRC, CR based on PET-CT was defined as complete MR in lymph nodes and ELS with a score of 1, 2, or 3 with or without residual mass, on 5PS where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake > mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions no evidence of FDG-avid disease in bone marrow. Bone marrow is normal by morphology; if indeterminate, IHC negative. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts) or after final dose of study treatment. Values have been rounded off to the nearest whole number.
Time Frame: 6-8 weeks after Cycle 6, Day 1 (cycle length is 21 days for DLBCL cohorts) or last dose of study drug (up to approximately 23 weeks)
Population: ITT population included all randomized participants in Arm H (Phase II NF Cohort) irrespective of whether or not they received the study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 64
percentage of participants | 42.2 [29.94 to 55.18]

8. Primary Outcome: Arm G (Phase II NF Cohort): Area Under Concentration-Time Curve (AUC) of Polatuzumab Vedotin (Lyophilized)
Description: Pharmacokinetic (PK) of three pola-related analytes: antibody conjugated monomethyl auristatin E (acMMAE), total antibody, and unconjugated MMAE were measured. The unit of measure for AUC is nanograms*day per milliliters.
Time Frame: Days 2, 8 and 15 of Cycle 1, Day 1 of Cycle 2 and 4, (each cycle is 21 days DLBCL cohorts) up to approximately 9 weeks
Population: PK population included all ITT participants in Arm G (Phase II NF Cohort) who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' is the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*day/mL
Arm/Group | Arm G (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 32
ng*day/mL
  acMMAE | 2880 (0.15)
  Total Antibody (Ab): number analyzed (Participants) | 0
  MMAE | 21.6 (45)

9. Primary Outcome: Arm G (Phase II NF Cohort): Maximum Concentration (Cmax) of Polatuzumab Vedotin (Lyophilized)
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Days 2, 8 and 15 of Cycle 1, Day 1 of Cycle 2 and 4,(cycle length is 21 days for DLBCL cohorts) up to approximately 9 weeks
Population: PK evaluable population included all the ITT participants in Arm G (Phase II NF Cohort) who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' is the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliters (ng/mL)
Arm/Group | Arm G (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 32
nanograms per milliliters (ng/mL)
  acMMAE | 724 (10)
  Total Ab: number analyzed (Participants) | 0
  MMAE | 2.01 (38)

10. Primary Outcome: Arm G (Phase II NF Cohort): Systemic Clearance (CL) of Polatuzumab Vedotin (Lyophilized)
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured. Unit of measure for CL is milliliters per day per kilograms (mL/day/kg)
Time Frame: Days 2, 8 and 15 of Cycle 1, Day 1 of Cycle 2 and 4, (cycle length is 21 days for DLBCL cohorts) up to approximately 9 weeks
Population: As pre-specified in the protocol the analysis of this outcome measure (OM) was based on sponsor's discretion however, sponsor opted to not collect data for this OM.
Arm/Group | Arm G (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 0

11. Primary Outcome: Arm G (Phase II NF Cohort): Steady-State Volume of Distribution (Vss) of Polatuzumab Vedotin (Lyophilized)
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Days 2, 8 and 15 of Cycle 1, Day 1 of Cycle 2 and 4, Day (cycle length is 21 days for DLBCL cohorts) up to approximately 9 weeks
Population: As pre-specified in the protocol the analysis of this OM was based on sponsor's discretion however, sponsor opted to not collect data for this OM.
Arm/Group | Arm G (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 0

12. Secondary Outcome: Phase II: Percentage of Participants With AEs
Description: as for outcome 2
Time Frame: From the study start up to the end of the study (up to approximately 84 months)
Population: Safety population consisted of all ITT participants from Phase II who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Groups:
- Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL: Participants with DLBCL received pola, 1.8 mg/kg, as IV infusion on Day 2 of Cycle 1 (each cycle is 21 days), and thereafter on Day 1 of Cycles 2 to 6. Participants also received bendamustine 90 mg/m^2, as IV infusion on Days 2 and 3 of Cycle 1, and thereafter on Days 1 and 2 of Cycles 2 to 6 and obinutuzumab 1000 mg, as IV infusion on Days 1, 8, and 15 of Cycle 1 and on Day 1 of Cycles 2 to 6 in combination with pola.
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 38 | 41 | 39 | 39 | 20 | 20 | 106
percentage of participants | 100 | 100 | 100 | 97.4 | 100 | 100 | 99.1

13. Secondary Outcome: Arms A and C (Phase II): Percentage of Participants With Treatment Emergent ADAs to Polatuzumab Vedotin
Description: The number of participants with positive results for ADA against pola at Baseline and at any of the post-baseline assessment time-points were reported. Participants positive at any post-baseline time points were post-baseline evaluable participants determined to have "Treatment-induced ADAs" or "Treatment-enhanced ADA" during the study period. Treatment-induced ADA = negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at baseline who has one or more post-baseline titer results that are at least 0.60 t.u. greater than the baseline titer result. Treatment emergent ADA is the sum of treatment-induced ADAs and treatment enhanced ADAs. Values have been rounded off to the nearest whole number.
Time Frame: Baseline to approximately Month 24
Population: Safety population consisted of all ITT participants from Arms A and C (Phase II) who received at least one dose of study medication. 'Overall Number Analyzed' is the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL
Number analyzed (Participants) | 38 | 36
percentage of participants
  Baseline Prevalence of ADAs: number analyzed (Participants) | 37 | 36
  Baseline Prevalence of ADAs | 0 | 0
  Post-Baseline Incidence of ADAs: number analyzed (Participants) | 38 | 35
  Post-Baseline Incidence of ADAs | 7.9 | 2.9

14. Secondary Outcome: Arms E and F (Phase II): Percentage of Participants With Treatment Emergent ADAs to Polatuzumab Vedotin and Obinutuzumab
Description: as for outcome 4
Time Frame: Baseline to approximately Month 24
Population: Safety population consisted of all ITT participants from Arms E and F (Phase II) who received at least one dose of study medication. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL
Number analyzed (Participants) | 20 | 20
percentage of participants
  Baseline Prevalence of ADAs to Polatuzumab: number analyzed (Participants) | 19 | 18
  Baseline Prevalence of ADAs to Polatuzumab | 0 | 0
  Post-Baseline Incidence of ADAs to Polatuzumab: number analyzed (Participants) | 19 | 18
  Post-Baseline Incidence of ADAs to Polatuzumab | 5.3 | 5.6
  Baseline Prevalence of ADAs to Obinutuzumab | 0 | 0
  Post-Baseline Incidence of ADAs to Obinutuzumab: number analyzed (Participants) | 19 | 18
  Post-Baseline Incidence of ADAs to Obinutuzumab | 0 | 0

15. Secondary Outcome: Phase II: Percentage of Participants With CR at PRA Based on PET-CT as Determined by the Investigator
Description: CR was assessed by investigator at PRA according to MLRC. Per MLRC, CR based on PET-CT was defined as complete MR in lymph nodes and ELS with a score of 1, 2, or 3 with or without residual mass, on 5PS where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake > mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions no evidence of FDG-avid disease in bone marrow. Bone marrow is normal by morphology; if indeterminate, IHC negative. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts and 28 days for FL cohorts) or after final dose of study treatment. As pre-specified in the protocol data reported is combined for Arms G and H. Values have been rounded off to the nearest whole number.
Time Frame: 6 to 8 weeks after Cycle 6 Day 1 (cycle length 21 days for DLBCL cohorts and 28 days for FL cohorts) or last dose of study drug (up to approximately 28 weeks)
Population: ITT population included all randomized participants in Phase II irrespective of whether or not they received the study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 39 | 41 | 40 | 40 | 20 | 21 | 106
percentage of participants | 64.1 [47.18 to 78.80] | 63.4 [46.94 to 77.88] | 42.5 [27.04 to 59.11] | 15.0 [5.71 to 29.84] | 65.0 [40.78 to 84.61] | 33.3 [14.59 to 56.97] | 36.8 [27.63 to 46.71]
Statistical Analysis 1: Comparison: Arm A (Phase II Randomization): Pola+BR in FL vs Arm B (Phase II Randomization): BR in FL; Test type: Superiority; p = 0.8817, Cochran-Mantel-Haenszel; Difference in Response Rates = 0.69, 95% CI 2-sided [-19.68 to 20.86]
Statistical Analysis 2: Comparison: Arm C (Phase II Randomization): Pola+BR in DLBCL vs Arm D (Phase II Randomization): BR in DLBCL; Test type: Superiority; p = 0.0061, Cochran-Mantel-Haenszel; Difference in Response Rates = 27.50, 95% CI 2-sided [7.66 to 44.74]

16. Secondary Outcome: Phase II Expansion Cohorts and Arm G (Phase II NF Cohort): Percentage of Participants With CR at PRA Based on PET-CT as Determined by the IRC
Description: CR was assessed by IRC at PRA according to MLRC. Per MLRC, CR based on PET-CT was defined as complete MR in lymph nodes and ELS with a score of 1, 2, or 3 with or without residual mass, on 5PS where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake > mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions no evidence of FDG-avid disease in bone marrow. Bone marrow is normal by morphology; if indeterminate, IHC negative. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts and 28 days for FL cohorts) or after final dose of study treatment. Values have been rounded off to the nearest whole number.
Time Frame: as for outcome 15
Population: ITT population included all randomized participants in Phase II Expansion Cohorts and Arm G (Phase II NF Cohort) irrespective of whether or not they received the study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm G (Phase II Expansion): Pola+BR in DLBCL: Participants with DLBCL received pola (lyophilized formulation), 1.8 mg/kg, as IV infusion on Day 2 of Cycle 1 (each cycle is 21 days), and thereafter on Day 1 of Cycles 2 to 6. Participants also received bendamustine 90 mg/m^2, as IV infusion on Days 2 and 3 of Cycle 1, and thereafter on Days 1 and 2 of Cycles 2 to 6 and rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1 to 6, in combination with pola.
Arm/Group | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G (Phase II Expansion): Pola+BR in DLBCL
Number analyzed (Participants) | 20 | 21 | 42
percentage of participants | 65.0 [40.78 to 84.61] | 33.3 [14.59 to 56.97] | 35.7 [21.55 to 51.97]

17. Secondary Outcome: Phase II: Percentage of Participants With Objective Response (OR) at PRA Based on PET-CT as Determined by Investigator
Description: OR at PRA was defined as the percentage of participants with CR or PR at the PRA, as assessed by the investigator according to MLRC. Per MLRC, CR based on PET-CT complete MR in lymph nodes and ELS with a score of 1, 2, or 3 with or without residual mass on 5PS, where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions; no new lesions and no evidence of FDG-avid disease in bone marrow, normal by morphology; if indeterminate, IHC negative. PR based on PET-CT was defined as partial MR in lymph nodes and ELS with a score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size at interim, residual uptake higher than uptake in normal bone marrow but reduced compared with baseline (diffuse uptake compatible with reactive changes from chemotherapy allowed).
Time Frame: 6 to 8 weeks after Cycle 6 Day 1 (cycle length 21 for DLBCL cohorts and 28 days for FL cohorts) or last dose of study drug (up to approximately 28 weeks)
Population: ITT population included all randomized participants in Phase II irrespective of whether or not they received the study treatment. As pre-specified in the protocol data reported is combined for Arms G and H. Values have been rounded off to the nearest whole number.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 39 | 41 | 40 | 40 | 20 | 21 | 106
percentage of participants | 79.5 [63.54 to 90.70] | 80.5 [63.13 to 91.18] | 47.5 [31.51 to 63.87] | 17.5 [7.34 to 32.78] | 85.0 [62.11 to 96.79] | 33.3 [14.59 to 56.97] | 42.5 [32.91 to 52.43]
Statistical Analysis 1: Comparison: Arm A (Phase II Randomization): Pola+BR in FL vs Arm B (Phase II Randomization): BR in FL; Test type: Superiority; p = 0.9523, Cochran-Mantel-Haenszel; Difference in Response Rates = -1.00, 95% CI 2-sided [-18.66 to 16.46]
Statistical Analysis 2: Comparison: Arm C (Phase II Randomization): Pola+BR in DLBCL vs Arm D (Phase II Randomization): BR in DLBCL; Test type: Superiority; p = 0.0036, Cochran-Mantel-Haenszel; Difference in Response Rates = 30.00, 95% CI 2-sided [9.48 to 47.37]

18. Secondary Outcome: Phase II: Percentage of Participants With OR at PRA Based on PET-CT as Determined by IRC
Description: OR at PRA was defined as the percentage of participants with CR or PR at the PRA, as assessed by the IRC according to MLRC. Per MLRC, CR based on PET-CT= complete MR in lymph nodes and ELS with a score of 1, 2, or 3 with or without residual mass on 5PS, where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions; no new lesions and no evidence of FDG-avid disease in bone marrow. Bone marrow normal by morphology; if indeterminate, IHC negative. PR based on PET-CT was defined as partial MR in lymph nodes and ELS with a score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size at interim, residual uptake higher than uptake in normal bone marrow but reduced compared with baseline (diffuse uptake compatible with reactive changes from chemotherapy allowed).
Time Frame: as for outcome 6
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 39 | 41 | 40 | 40 | 20 | 21 | 106
percentage of participants | 76.9 [60.67 to 88.87] | 73.2 [57.06 to 85.78] | 42.5 [27.04 to 59.11] | 17.5 [7.34 to 32.78] | 85.0 [62.11 to 96.79] | 38.1 [18.11 to 61.56] | 43.4 [33.80 to 53.37]
Statistical Analysis 1: Comparison: Arm A (Phase II Randomization): Pola+BR in FL vs Arm B (Phase II Randomization): BR in FL; Test type: Superiority; p = 0.6574, Cochran-Mantel-Haenszel; Difference in Response Rates = 3.75, 95% CI 2-sided [-15.14 to 22.11]
Statistical Analysis 2: Comparison: Arm C (Phase II Randomization): Pola+BR in DLBCL vs Arm D (Phase II Randomization): BR in DLBCL; Test type: Superiority; p = 0.0128, Cochran-Mantel-Haenszel; Difference in Response Rates = 25.00, 95% CI 2-sided [4.89 to 42.63]

19. Secondary Outcome: Phase II: Percentage of Participants With CR at PRA Based on CT Only as Determined by Investigator
Description: CR was determined by investigator at PRA according to the MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 centimetres (cm) in in longest transverse diameter (LDi) and no ELS of disease organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, IHC negative. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts and 28 days for FL cohorts). As pre-specified in the protocol data reported is combined for Arms G and H. Values have been rounded off to the nearest whole number.
Time Frame: as for outcome 6
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 39 | 41 | 40 | 40 | 20 | 21 | 106
percentage of participants | 46.2 [30.09 to 62.82] | 19.5 [8.82 to 34.87] | 20.0 [9.05 to 35.65] | 5.0 [0.61 to 16.92] | 20.0 [5.73 to 43.66] | 14.3 [3.05 to 36.34] | 14.2 [8.14 to 22.26]

20. Secondary Outcome: Phase II: Percentage of Participants With CR at PRA Based on CT Only as Determined by IRC
Description: CR was determined by IRC a at PRA according to the MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, IHC negative. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts and 28 days for FL cohorts). As pre-specified in the protocol data reported is combined for Arms G and H. Values have been rounded off to the nearest whole number.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 39 | 41 | 40 | 40 | 20 | 20 | 106
percentage of participants | 41.0 [25.57 to 57.90] | 36.6 [22.12 to 53.06] | 22.5 [10.84 to 38.45] | 2.5 [0.06 to 13.16] | 50.0 [27.20 to 72.80] | 23.8 [8.22 to 47.17] | 17.9 [11.15 to 26.57]

21. Secondary Outcome: Phase II: Percentage of Participants With OR at PRA Based on CT Only as Determined by Investigator
Description: OR at PRA was defined as the percentage of participants with CR or PR at the PRA, as assessed by the investigator based on MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease organ enlargement regressing to normal; no new lesions; bone marrow normal by morphology, if indeterminate, IHC negative. PR per CT only was defined as partial remission in lymph nodes and ELS with ≥50% decrease in sum of the products of greatest diameters (SPD) of up to 6 target measurable lymph nodes and extranodal sites, absent/normal/regressed but with no increase in non-measured lesions, spleen regressing by ≥50% in length beyond normal it, no new sites of lesions. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts and 28 days for FL cohorts).
Time Frame: as for outcome 6
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 39 | 41 | 40 | 40 | 20 | 21 | 106
percentage of participants | 79.5 [63.54 to 90.70] | 75.6 [59.70 to 87.64] | 45.0 [29.26 to 61.51] | 15.0 [5.71 to 29.84] | 80.0 [56.34 to 94.27] | 33.3 [14.59 to 56.97] | 42.5 [32.91 to 52.43]
Statistical Analysis 1: Comparison: Arm A (Phase II Randomization): Pola+BR in FL vs Arm B (Phase II Randomization): BR in FL; Test type: Superiority; p = 0.6225, Cochran-Mantel-Haenszel; Difference in Response Rates = 3.88, 95% CI 2-sided [-14.49 to 21.72]
Statistical Analysis 2: Comparison: Arm C (Phase II Randomization): Pola+BR in DLBCL vs Arm D (Phase II Randomization): BR in DLBCL; Test type: Superiority; p = 0.0032, Cochran-Mantel-Haenszel; Difference in Response Rates = 30.00, 95% CI 2-sided [9.94 to 47.12]

22. Secondary Outcome: Phase II: Percentage of Participants With OR at PRA Based on CT Only as Determined by IRC
Description: OR at PRA was defined as the percentage of participants with CR or PR at the PRA, as assessed by the IRC based on MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease organ enlargement regressing to normal; no new lesions; bone marrow normal by morphology, if indeterminate, IHC negative. PR per CT only was defined as partial remission in lymph nodes and ELS with ≥50% decrease SPD of up to 6 target measurable lymph nodes and extranodal sites, absent/normal/regressed but with no increase in non-measured lesions, spleen regressing by ≥50% in length beyond normal it, no new sites of lesions. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts and 28 days for FL cohorts).
Time Frame: as for outcome 6
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 39 | 41 | 40 | 40 | 20 | 21 | 106
percentage of participants | 74.4 [57.87 to 86.96] | 80.5 [65.13 to 91.18] | 40.0 [24.86 to 56.67] | 15.0 [5.71 to 29.84] | 80.0 [56.34 to 94.27] | 38.1 [18.11 to 61.56] | 41.5 [32.02 to 51.49]
Statistical Analysis 1: Comparison: Arm A (Phase II Randomization): Pola+BR in FL vs Arm B (Phase II Randomization): BR in FL; Test type: Superiority; p = 0.4835, Cochran-Mantel-Haenszel; Difference in Response Rates = -6.13, 95% CI 2-sided [-24.14 to 12.12]
Statistical Analysis 2: Comparison: Arm C (Phase II Randomization): Pola+BR in DLBCL vs Arm D (Phase II Randomization): BR in DLBCL; Test type: Superiority; p = 0.0096, Cochran-Mantel-Haenszel; Difference in Response Rates = 25.00, 95% CI 2-sided [5.39 to 42.33]

23. Secondary Outcome: Phase II: Percentage of Participants With Best Objective Response (BOR) Based on PET-CT or CT Only as Determined by the Investigator
Description: BOR=CR/PR per PET-CT/CT per MLRC.CR per PET-CT=complete MR in LN & ELS, score=1, 2,3 with/without a residual mass on 5-PS; 1=no uptake(UT) above background;2=UT≤mediastinum;3=UT>mediastinum but ≤liver;4=UT moderately>liver;5=UT markedly higher than liver &/or new lesions;no evidence of FDG-avid disease, bone marrow morphology=normal;if indeterminate, is IHC negative.PR per PET-CT=partial MR in LN & ELS, score=4 or 5, reduced UT than baseline (BL) & residual mass of any size;residual UT>UT in normal marrow but reduced than BL.CR per CT=complete radiologic response with target nodes/nodal masses regressed to ≤1.5cm in LDi & no ELS of disease, absences of non-measured lesion;organ enlargement regressed to normal;no new lesions;bone marrow= normal;if indeterminate, is IHC negative.PR per CT=≥50% decrease in SPD of up to 6 target nodes & extranodal sites;non-measured lesions=absent/normal/regressed/no increase;spleen=regressed by ≥50% in length beyond normal, no new lesions.
Time Frame: Up to every 6 months until disease progression, withdrawal or study completion (up to approximately 84 months)
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 39 | 41 | 40 | 40 | 20 | 21 | 106
percentage of participants | 89.7 [75.78 to 97.13] | 90.2 [76.87 to 97.28] | 70.0 [53.47 to 83.44] | 32.5 [18.57 to 49.13] | 90.0 [68.30 to 98.77] | 52.4 [29.78 to 74.29] | 62.3 [52.33 to 71.50]
Statistical Analysis 1: Comparison: Arm A (Phase II Randomization): Pola+BR in FL vs Arm B (Phase II Randomization): BR in FL; Test type: Superiority; p = 0.9390, Cochran-Mantel-Haenszel; Difference in Response Rates = -0.50, 95% CI 2-sided [-15.07 to 13.71]
Statistical Analysis 2: Comparison: Arm C (Phase II Randomization): Pola+BR in DLBCL vs Arm D (Phase II Randomization): BR in DLBCL; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel; Difference in Response Rates = 37.50, 95% CI 2-sided [15.64 to 54.71]

24. Secondary Outcome: DLBCL Cohorts: Percentage of Participants With BOR Based PET-CT or CT Only as Determined by IRC
Description: as for outcome 23
Time Frame: Up to every 6 months until disease progression, withdrawal or study completion (up to approximately 84 months)
Population: ITT population included all randomized participants in DLBCL Cohorts irrespective of whether or not they received the study treatment. As pre-specified in the protocol data reported is combined for Arms G and H. Values have been rounded off to the nearest whole number.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 40 | 40 | 21 | 106
percentage of participants | 62.5 [45.80 to 77.27] | 25.0 [12.69 to 41.20] | 42.9 [21.82 to 65.98] | 57.5 [47.57 to 67.09]
Statistical Analysis 1: Comparison: Arm C (Phase II Randomization): Pola+BR in DLBCL vs Arm D (Phase II Randomization): BR in DLBCL; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel; Difference in Response Rates = 37.50, 95% CI 2-sided [15.82 to 54.62]

25. Secondary Outcome: DLBCL Cohorts: Duration of Response (DOR) Based on PET-CT or CT Only as Determined by the Investigator
Description: DOR=first occurrence of CR/PR to disease progression/relapse/death per PET-CT/CT, per investigator per MLRC.CR per PET-CT=score 1/2/3 with/without a residual mass on 5-PS for LN and ELS;1=no UT> background; 2=UT≤mediastinum;3=UT>mediastinum but ≤liver;4=UT moderately>liver;5=UT>than liver &/or new lesions;bone marrow morphology=no evidence of FDG-avid disease, normal;if indeterminate IHC negative.PR per PET-CT=score of 4/5 with reduced UT compared to BL & residual mass of any size at interim for LN & ELS;residual UT>UT in normal bone marrow but<than BL. CR per CT=target nodes/nodal masses regressed to ≤1.5cm in LDi no ELS of disease for LN & ELS, no non-measured lesion, organ enlargement regressed to normal; bone marrow=normal morphology; if indeterminate, IHC negative. PR per CT= ≥50% decrease SPD of 6 target measurable LN and extranodal sites, absent/normal/regressed but no increase in non-measured lesions, spleen ≥50% in length beyond normal involvement, no new sites of lesions.
Time Frame: From the date of the first occurrence of a documented CR or PR to the date of disease progression, relapse, or death from any cause whichever occur first (up to approximately 84 months)
Population: ITT population included all randomized participants in DLBCL Cohorts irrespective of whether or not they received the study treatment. As pre-specified in the protocol data reported is combined for Arms G and H. 'Overall Number Analyzed' are the number of participants with data available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 28 | 13 | 11 | 66
months | 12.665 [5.782 to 27.926] | 4.074 [2.563 to 12.682] | 16.099 [2.825 to 27.860] | 11.335 [6.242 to 16.197]
Statistical Analysis 1: Comparison: Arm C (Phase II Randomization): Pola+BR in DLBCL vs Arm D (Phase II Randomization): BR in DLBCL; Test type: Superiority; p = 0.0245, Log Rank; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.19 to 0.91]

26. Secondary Outcome: DLBCL Cohorts: DOR Based on PET-CT or CT Only as Determined by the IRC
Description: DOR=first occurrence of CR/PR to disease progression/relapse/death per PET-CT/CT, per IRC per MLRC.CR per PET-CT=score 1/2/3 with/without a residual mass on 5-PS for LN and ELS;1=no UT> background; 2=UT≤mediastinum;3=UT>mediastinum but ≤liver;4=UT moderately>liver;5=UT>than liver &/or new lesions;bone marrow morphology=no evidence of FDG-avid disease, normal;if indeterminate IHC negative.PR per PET-CT=score of 4/5 with reduced UT compared to BL & residual mass of any size at interim for LN & ELS;residual UT>UT in normal bone marrow but<than BL. CR per CT=target nodes/nodal masses regressed to ≤1.5cm in LDi no ELS of disease for LN & ELS, no non-measured lesion, organ enlargement regressed to normal; bone marrow=normal morphology; if indeterminate, IHC negative. PR per CT= ≥50% decrease SPD of 6 target measurable LN and extranodal sites, absent/normal/regressed but no increase in non-measured lesions, spleen ≥50% in length beyond normal involvement, no new sites of lesions.
Time Frame: as for outcome 25
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 25 | 10 | 9 | 61
months | 10.908 [5.684 to 40.674] | 10.645 [3.975 to 19.647] | 25.758 [9.692 to 46.752] | 13.437 [8.641 to 20.041]
Statistical Analysis 1: Comparison: Arm C (Phase II Randomization): Pola+BR in DLBCL vs Arm D (Phase II Randomization): BR in DLBCL; Test type: Superiority; p = 0.2451, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.25 to 1.43]

27. Secondary Outcome: DLBCL Cohorts: Progression Free Survival (PFS) Based on PET-CT or CT Only as Determined by the Investigator
Description: PFS was defined as the time randomization or from first study treatment (for obinuzumab arms) to the first occurrence of disease progression, relapse or death, from any cause based on PET-CT or CT only, as determined by the investigators assessment. As pre-specified in the protocol data reported is combined for Arms G and H.
Time Frame: From the date of randomization or first treatment to the first occurrence of progression or relapse, or death from any cause (up to approximately 84 months)
Population: ITT population included all randomized participants in DLBCL Cohorts irrespective of whether or not they received the study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 40 | 40 | 21 | 106
months | 7.491 [4.928 to 16.953] | 2.037 [1.544 to 3.713] | 5.125 [2.103 to 18.234] | 5.881 [4.764 to 7.524]
Statistical Analysis 1: Comparison: Arm C (Phase II Randomization): Pola+BR in DLBCL vs Arm D (Phase II Randomization): BR in DLBCL; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.20 to 0.56]

28. Secondary Outcome: DLBCL Cohorts: PFS Based on PET-CT or CT Only as Determined by the IRC
Description: PFS was defined as the time randomization or from first study treatment (for obinuzumab arms) to the first occurrence of disease progression, relapse or death, from any cause based on PET-CT or CT only, as determined by the IRC assessment. As pre-specified in the protocol data reported is combined for Arms G and H.
Time Frame: as for outcome 27
Population: as for outcome 27
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 40 | 40 | 21 | 106
months | 9.248 [6.045 to 13.930] | 3.713 [2.070 to 4.534] | 5.848 [2.103 to 11.893] | 6.965 [5.092 to 9.823]
Statistical Analysis 1: Comparison: Arm C (Phase II Randomization): Pola+BR in DLBCL vs Arm D (Phase II Randomization): BR in DLBCL; Test type: Superiority; p = 0.0003, Log Rank; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.23 to 0.66]

29. Secondary Outcome: Phase II NF Cohort: Percentage of Participants With CR at PRA Based on PET-CT as Determined by the Investigator
Description: CR was assessed by Investigator at PRA according to MLRC. Per MLRC, CR based on PET-CT was defined as complete MR in lymph nodes and ELS with a score of 1, 2, or 3 with or without residual mass, on 5PS where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake > mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions no evidence of FDG-avid disease in bone marrow. Bone marrow is normal by morphology; if indeterminate, IHC negative. As pre-specified in the protocol data reported is combined for Arms G and H. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts) or after final dose of study treatment. Values have been rounded off to the nearest whole number.
Time Frame: 6 to 8 weeks after Cycle 6 Day 1 (cycle length 21 days for DLBCL cohorts) or last dose of study drug (up to approximately 23 weeks)
Population: ITT population included all randomized participants in Phase II NF Cohort irrespective of whether or not they received the study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 106
percentage of participants | 36.8 [27.63 to 46.71]

30. Secondary Outcome: Phase II NF Cohort: Percentage of Participants With OR at PRA Based on PET-CT as Determined by Investigator
Description: OR at PRA was defined as the percentage of participants with CR or PR at the PRA, as assessed by the investigator according to MLRC. Per MLRC, CR based on PET-CT= complete MR in lymph nodes and ELS with a score of 1, 2, or 3 with or without residual mass on 5PS, where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake mediastinum but ≤ liver; 4=uptake moderately>liver; 5=uptake markedly higher than liver and/or new lesions ; no new lesions and no evidence of FDG-avid disease in bone marrow, normal by morphology; if indeterminate, IHC negative. PR based on PET-CT was defined as partial MR in lymph nodes and ELS with a score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size at interim, residual uptake higher than uptake in normal bone marrow but reduced compared with baseline (diffuse uptake compatible with reactive changes from chemotherapy allowed).
Time Frame: 6 to 8 weeks after Cycle 6 Day 1 (cycle length is 21 days for DLBCL cohorts) or last dose of study drug (up to approximately 23 weeks)
Population: ITT population included all randomized participants in Phase II NF Cohort irrespective of whether or not they received the study treatment. As pre-specified in the protocol data reported is combined for Arms G and H. Values have been rounded off to the nearest whole number.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 106
percentage of participants | 42.5 [32.91 to 52.43]

31. Secondary Outcome: Phase II NF Cohort: Percentage of Participants With OR at PRA Based on PET-CT as Determined by IRC
Description: OR at PRA was defined as the percentage of participants with CR or PR at the PRA, as assessed by the IRC according to MLRC. Per MLRC, CR based on PET-CT= complete MR in lymph nodes and ELS with a score of 1, 2, or 3 with or without residual mass on 5PS, where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions ; no new lesions and no evidence of FDG-avid disease in bone marrow, bone marrow normal by morphology; if indeterminate, IHC negative. PR based on PET-CT was defined as partial MR in lymph nodes and ELS with a score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size at interim, residual uptake higher than uptake in normal bone marrow but reduced compared with baseline (diffuse uptake compatible with reactive changes from chemotherapy allowed).
Time Frame: as for outcome 30
Population: as for outcome 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 106
percentage of participants | 43.4 [33.80 to 53.37]

32. Secondary Outcome: Phase II NF Cohorts: Percentage of Participants With BOR Based on PET-CT or CT Only as Determined by the Investigator
Description: BOR=CR/PR per PET-CT/CT per MLRC. CR per PET-CT=complete MR in lymph nodes & ELS, score=1, 2,3 with/without a residual mass on 5-PS; 1=no UT above background; 2=UT≤mediastinum;3=UT>mediastinum but ≤liver;4=UT moderately>liver;5=UT markedly higher than liver &/or new lesions;no evidence of FDG-avid disease, bone marrow morphology=normal;if indeterminate, is IHC negative.PR per PET-CT=partial MR in lymph nodes & ELS, score=4 or 5, reduced UT than BL & residual mass of any size;residual UT>UT in normal marrow but reduced than BL.CR per CT=complete radiologic response with target nodes/nodal masses regressed to ≤1.5cm in LDi & no ELS of disease, absences of non-measured lesion;organ enlargement regressed to normal;no new lesions;bone marrow= normal;if indeterminate, is IHC negative.PR per CT=≥50% decrease in SPD of up to 6 target nodes & extranodal sites;non-measured lesions=absent/normal/regressed/no increase;spleen=regressed by ≥50% in length beyond normal, no new lesions.
Time Frame: Up to every 6 months until disease progression, withdrawal or study completion (from Month 37 to Month 84 [up to approximately 47 months])
Population: as for outcome 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 106
percentage of participants | 62.3 [52.33 to 71.50]

33. Secondary Outcome: Phase II NF Cohorts: Percentage of Participants With BOR Based on PET-CT or CT Only as Determined by the IRC
Description: as for outcome 32
Time Frame: as for outcome 32
Population: as for outcome 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 106
percentage of participants | 57.5 [47.57 to 67.09]

34. Secondary Outcome: Phase II NF Cohort: DOR Based on PET-CT or CT Only as Determined by the Investigator
Description: as for outcome 25
Time Frame: From the date of the first occurrence of a documented CR or PR to the date of disease progression, relapse, or death from any cause whichever occur first (from Month 37 to Month 84 [up to approximately 47 months])
Population: ITT population included all randomized participants in Phase II NF Cohort irrespective of whether or not they received the study treatment. As pre-specified in the protocol data reported is combined for Arms G and H. 'Overall Number Analyzed' are the number of participants with data available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 66
months | 11.335 [6.242 to 16.197]

35. Secondary Outcome: Phase II NF Cohort: DOR Based on PET-CT or CT Only as Determined by the IRC
Description: as for outcome 26
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 61
months | 13.437 [8.641 to 20.041]

36. Secondary Outcome: Phase II NF Cohort: PFS Based on PET-CT or CT Only as Determined by the Investigator
Description: PFS was defined as the time from randomization or from first study treatment (for obinuzumab arms) to the first occurrence of disease progression, relapse or death, from any cause based on PET-CT or CT only, as determined by the investigators assessment. As pre-specified in the protocol data reported is combined for Arms G and H.
Time Frame: From the date of randomization or first treatment to the first occurrence of progression or relapse, or death from any cause (from Month 37 to Month 84 [up to approximately 47 months])
Population: as for outcome 29
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 106
months | 5.881 [4.764 to 7.524]

37. Secondary Outcome: Phase II NF Cohort: PFS Based on PET-CT or CT Only as Determined by the IRC
Description: PFS was defined as the time from randomization or from first study treatment (for obinuzumab arms) to the first occurrence of disease progression, relapse or death, from any cause based on PET-CT or CT only, as determined by the IRC assessment. As pre-specified in the protocol data reported is combined for Arms G and H.
Time Frame: as for outcome 36
Population: as for outcome 29
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 106
months | 6.965 [5.092 to 9.823]

38. Secondary Outcome: Phase II NF Cohort: Event-Free Survival (EFS) Based on PET-CT or CT Only, as Determined by the Investigator
Description: EFS was defined as time from randomization to disease progression or relapse, as assessed by the investigator or death from any cause. As pre-specified in the protocol data reported is combined for Arms G and H.
Time Frame: From Month 37 to Month 84 (up to approximately 47 months)
Population: as for outcome 29
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 106
months | 5.092 [4.402 to 6.867]

39. Secondary Outcome: Phase II NF Cohorts: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization or first treatment (for obinutuzumab arms) to the date of death from any cause. As pre-specified in the protocol data reported is combined for Arms G and H.
Time Frame: From Month 37 to Month 84 (up to approximately 47 months)
Population: as for outcome 29
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 106
months | 12.320 [8.279 to 16.986]

40. Secondary Outcome: Arm G (Phase II NF Cohort): Percentage of Participants With CR at PRA Based on PET-CT as Determined by the IRC
Description: CR was assessed by IRC at PRA according to MLRC. Per MLRC, CR based on PET-CT was defined as complete MR in lymph nodes and ELS with a score of 1, 2, or 3 with or without residual mass, on 5PS where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake > mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions no evidence of FDG-avid disease in bone marrow. Bone marrow is normal by morphology; if indeterminate, IHC negative. As pre-specified in the protocol data reported is combined for Arms G and H. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts) or after final dose of study treatment. Values have been rounded off to the nearest whole number.
Time Frame: as for outcome 30
Population: ITT population included all randomized participants in Arm G (Phase II NF Cohort) irrespective of whether or not they received the study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm G (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 42
percentage of participants | 35.7 [21.55 to 51.97]

41. Secondary Outcome: Arm G (Phase II NF Cohort): Percentage of Participants With CR at PRA Based on CT Only as Determined by Investigator
Description: CR was determined by Investigator at PRA according to the MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, IHC negative. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts). Values have been rounded off to the nearest whole number.
Time Frame: as for outcome 30
Population: as for outcome 40
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm G (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 42
percentage of participants | 9.5 [2.66 to 22.62]

42. Secondary Outcome: Arm G (Phase II NF Cohort): Percentage of Participants With CR at PRA Based on CT Only as Determined by IRC
Description: CR was determined by IRC at PRA according to the MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, IHC negative. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts). Values have been rounded off to the nearest whole number.
Time Frame: as for outcome 30
Population: as for outcome 40
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm G (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 42
percentage of participants | 14.3 [5.43 to 28.54]

43. Secondary Outcome: Arm G (Phase II NF Cohort): Percentage of Participants With OR at PRA Based on CT Only as Determined by Investigator
Description: OR at PRA was defined as the percentage of participants with CR or PR at the PRA, as assessed by the investigator based on MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, IHC negative. PR per CT only was defined as partial remission in lymph nodes and ELS with ≥50% decrease in SPD of up to 6 target measurable lymph nodes and extranodal sites, absent/normal/regressed but with no increase in non-measured lesions, spleen regressing by ≥50% in length beyond normal it, no new sites of lesions. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts).
Time Frame: 6 to 8 weeks after Cycle 6 Day 1 (cycle length is 21 days for DLBCL cohorts) or last dose of study drug (up to 23 weeks)
Population: ITT population included all randomized participants in Arm G (Phase II NF Cohort) irrespective of whether or not they received the study treatment. Values have been rounded off to the nearest whole number.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm G (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 42
percentage of participants | 38.1 [23.57 to 54.36]

44. Secondary Outcome: Arm G (Phase II NF Cohort): Percentage of Participants With OR at PRA Based on CT Only as Determined by IRC
Description: OR at PRA was defined as the percentage of participants with CR or PR at the PRA, as assessed by the IRC based on MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, IHC negative. PR per CT only was defined as partial remission in lymph nodes and ELS with ≥50% decrease in SPD of up to 6 target measurable lymph nodes and extranodal sites, absent/normal/regressed but with no increase in non-measured lesions, spleen regressing by ≥50% in length beyond normal it, no new sites of lesions. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 21 days for DLBCL cohorts).
Time Frame: as for outcome 43
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm G (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 42
percentage of participants | 33.3 [19.57 to 49.55]

45. Secondary Outcome: Plasma Concentration of of Polatuzumab Vedotin Analyte: acMMAE
Description: PK of pola-related analyte acMMAE was measured. Cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts.
Time Frame: Cycle 1 Day 2: pre-dose and 30 minutes (min) post dose; Cycle 1 Days 8 and 15; Cycle 2 and 4 Day 1: pre-dose and 30 min post dose; unscheduled visits: pre-dose and 30 min post dose; study treatment completion (up to approximately 84 months)
Population: PK evaluable population included all the ITT participants in Phase Ib and Phase II who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL | Arm A (Phase II Randomization): Pola+BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 36 | 36 | 18 | 19
ng/mL
  Cycle 1 Day 2: Pre-dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 36 | 36 | 17 | 16
  Cycle 1 Day 2: Pre-dose | NA (NA) — The data is not evaluable as the samples were below lower limit of quantification (BLLQ). | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ.
  Cycle 1 Day 2: 30 min Post Dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 36 | 35 | 18 | 19
  Cycle 1 Day 2: 30 min Post Dose | 654 (29.3) | 617 (26.2) | 719 (26.7) | 718 (14.2) | 492 (241.6) | 643 (24.7) | 453 (682.8) | 472 (617.2)
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 6 | 6 | 6 | 0 | 0 | 0 | 0
  Cycle 1 Day 8 | 29.4 (5887.2) | 75.9 (40.8) | 90.7 (46.1) | 109 (48.2) |  |  |  |
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 6 | 5 | 6 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 | 12.2 (1626.9) | 25.4 (29.8) | 28.9 (48.6) | 34.4 (37.3) |  |  |  |
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 35 | 33 | 18 | 16
  Cycle 2 Day 1: Pre-dose | 3.21 (546.5) | 12.4 (47.9) | 8.75 (77.7) | 16.6 (25.6) | 4.72 (159.8) | 12.7 (120.5) | 9.05 (74.4) | 13.1 (45.2)
  Cycle 2 Day 1: 30 min Post Dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: 30 min Post Dose | 685 (22.0) | 683 (20.1) | 803 (20.1) | 834 (13.5) |  |  |  |
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 5 | 3 | 6 | 4 | 31 | 23 | 16 | 12
  Cycle 4 Day 1: Pre-dose | 12.2 (26.1) | 21.1 (46.7) | 15.3 (61.9) | 26.2 (22.1) | 11.2 (109.3) | 20.7 (46.4) | 15.2 (30.5) | 19.6 (30.5)
  Cycle 4 Day 1: 30 min Post Dose: number analyzed (Participants) | 5 | 3 | 6 | 4 | 29 | 23 | 17 | 12
  Cycle 4 Day 1: 30 min Post Dose | 748 (23.4) | 754 (14.4) | 734 (22.0) | 716 (13.7) | 689 (20.9) | 645 (21.4) | 829 (20.3) | 709 (10.1)
  Unscheduled Visit: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0
  Unscheduled Visit |  |  |  |  |  | 41.1 (49.4) | 53.0 (58.0) |
  Unscheduled Visit: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Unscheduled Visit: Pre-dose |  |  |  |  | 1.21 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 0.180 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  |
  Unscheduled Visit: 30 min Post Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Unscheduled Visit: 30 min Post Dose |  |  |  |  |  | 915 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  |
  Study Treatment Completion: number analyzed (Participants) | 0 | 0 | 1 | 0 | 28 | 27 | 14 | 8
  Study Treatment Completion |  |  | 18.7 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 10.7 (181.7) | 14.2 (95.7) | 14.9 (69.4) | 12.3 (109.4)

46. Secondary Outcome: Arm G+H (Phase II NF Cohorts): Plasma Concentration of of Polatuzumab Vedotin Analyte: acMMAE
Description: PK of one pola-related analytes: acMMAE was measured. Cycle length is 21 days for DLBCL cohorts. As pre-specified in the protocol data is reported combined for arms G+H.
Time Frame: Cycle 1 Day 2: post dose; Cycle 2 and 4 Day 1: pre-dose and post dose
Population: PK evaluable population included all the ITT participants in Arm G+H (Phase II NF Cohort) who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 102
ng/mL
  Cycle 1 Day 2: Post Dose | 653 (237)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 94
  Cycle 2 Day 1: Pre-dose | 14.6 (8.66)
  Cycle 2 Day 1: Post Dose: number analyzed (Participants) | 92
  Cycle 2 Day 1: Post Dose | 667 (155)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 61
  Cycle 4 Day 1: Pre-dose | 23.2 (8.59)
  Cycle 4 Day 1: Post Dose: number analyzed (Participants) | 60
  Cycle 4 Day 1: Post Dose | 659 (156)

47. Secondary Outcome: Serum Concentration of of Polatuzumab Vedotin Analyte: Total Ab
Description: PK of pola-related analyte Total Ab was measured. Cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts.
Time Frame: Cycle 1 Days 2: pre-dose & 30 min post dose; Cycle 1 Days 8 & 15; Cycle 2 and 4 Day 1 and unscheduled visits: pre-dose & 30 min post dose; Follow up at Day 1: Months 3, 6, 12, 18 & 24; study treatment completion visit (up to approx. 84 months)
Population: PK evaluable population included all the ITT participants Phase Ib and Phase II who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: grams per milliliters (g/mL)
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL | Arm A (Phase II Randomization): Pola+BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 36 | 36 | 18 | 19
grams per milliliters (g/mL)
  Cycle 1 Day 2: Pre-dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 36 | 36 | 17 | 18
  Cycle 1 Day 2: Pre-dose | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ.
  Cycle 1 Day 2: 30 min Post Dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 36 | 35 | 18 | 19
  Cycle 1 Day 2: 30 min Post Dose | 33.2 (28.4) | 36.6 (25.4) | 37.5 (29.1) | 34.3 (20.3) | 35.4 (27.7) | 34.6 (26.2) | 32.4 (22.8) | 38.3 (20.3)
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 6 | 6 | 6 | 0 | 0 | 0 | 0
  Cycle 1 Day 8 | 3.43 (4393.4) | 9.01 (43.7) | 10.2 (39.3) | 10.0 (31.9) |  |  |  |
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 6 | 6 | 6 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 | 1.83 (1784.3) | 4.26 (35.3) | 4.61 (40.6) | 5.22 (28.4) |  |  |  |
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 36 | 33 | 18 | 16
  Cycle 2 Day 1: Pre-dose | 0.696 (941.2) | 2.31 (54.2) | 2.20 (76.1) | 3.70 (27.4) | 1.23 (203.1) | 2.48 (137.6) | 2.20 (100.6) | 2.83 (41.8)
  Cycle 2 Day 1: 30 min Post Dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: 30 min Post Dose | 35.8 (25.9) | 39.5 (28.3) | 43.4 (31.1) | 42.2 (22.9) |  |  |  |
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 5 | 3 | 6 | 4 | 32 | 23 | 16 | 12
  Cycle 4 Day 1: Pre-dose | 3.44 (30.5) | 5.03 (59.0) | 4.61 (62.2) | 6.26 (18.3) | 3.61 (97.8) | 5.72 (39.9) | 4.82 (20.8) | 5.03 (29.3)
  Cycle 4 Day 1: 30 min Post Dose: number analyzed (Participants) | 5 | 3 | 6 | 4 | 31 | 23 | 17 | 12
  Cycle 4 Day 1: 30 min Post Dose | 40.2 (27.2) | 44.6 (11.0) | 43.0 (25.8) | 47.1 (24.2) | 44.8 (24.3) | 40.6 (20.6) | 55.0 (21.3) | 37.5 (11.6)
  Follow up on Month 3, Day 1: number analyzed (Participants) | 5 | 3 | 5 | 2 | 23 | 18 | 15 | 8
  Follow up on Month 3, Day 1 | 0.164 (51.9) | 0.771 (193.4) | 0.910 (82.8) | 0.394 (27.1) | 0.265 (209.9) | 0.316 (266.2) | 0.489 (174.2) | 0.543 (126.7)
  Follow up on Month 6, Day 1: number analyzed (Participants) | 5 | 3 | 5 | 2 | 21 | 12 | 10 | 7
  Follow up on Month 6, Day 1 | 0.0250 (0.0) | 0.0788 (230.0) | 0.219 (96.6) | 0.104 (18.5) | 0.0539 (145.7) | 0.0564 (195.7) | 0.0920 (123.5) | 0.150 (206.6)
  Follow up on Month 12, Day 1: number analyzed (Participants) | 4 | 3 | 4 | 3 | 13 | 9 | 6 | 3
  Follow up on Month 12, Day 1 | 0.0250 (0.0) | 0.0250 (0.0) | 0.0298 (35.9) | 0.0250 (0.0) | 0.0250 (0.0) | 0.0301 (60.6) | 0.0250 (0.0) | 0.0250 (0.0)
  Follow up on Month 18, Day 1: number analyzed (Participants) | 2 | 3 | 2 | 2 | 2 | 0 | 3 | 3
  Follow up on Month 18, Day 1 | 0.0250 (0.0) | 0.0250 (0.0) | 0.0250 (0.0) | 0.0250 (0.0) | 0.0250 (0.0) |  | 0.0250 (0.0) | 0.0250 (0.0)
  Follow up on Month 24, Day 1: number analyzed (Participants) | 2 | 3 | 1 | 1 | 0 | 0 | 0 | 1
  Follow up on Month 24, Day 1 | 0.0250 (0.0) | 0.0250 (0.0) | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated.. |  |  |  | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated.
  Unscheduled Visit: number analyzed (Participants) | 3 | 2 | 0 | 1 | 0 | 4 | 3 | 0
  Unscheduled Visit | 0.0250 (0.0) | 0.0250 (0.0) |  | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 1.65 (5419.8) | 1.23 (30267.8) |
  Unscheduled Visit: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Unscheduled Visit: Pre-dose |  |  |  |  | 0.279 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  |
  Unscheduled Visit: 30 min Post Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Unscheduled Visit: 30 min Post Dose |  |  |  |  |  | 42.0 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  |
  Study Treatment Completion Visit: number analyzed (Participants) | 0 | 0 | 1 | 0 | 27 | 27 | 14 | 8
  Study Treatment Completion Visit |  |  | 5.34 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 3.34 (180.5) | 4.33 (69.4) | 4.57 (57.2) | 3.23 (79.3)

48. Secondary Outcome: Arm G+H (Phase II NF Cohorts): Plasma Concentration of Polatuzumab Vedotin Analyte: Total Ab
Description: PK of pola-related analyte: Total Ab was measured. Cycle length is 21 days for DLBCL cohorts. As pre-specified in the protocol data is reported combined for arms G+H.
Time Frame: Cycle 1 Day 2: post dose; Cycle 2 and 4 Day 1: pre-dose and post dose
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 103
ng/mL
  Cycle 1 Day 2: Post Dose | 33.9 (11.7)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 94
  Cycle 2 Day 1: Pre-dose | 3.27 (4.37)
  Cycle 2 Day 1: Post Dose: number analyzed (Participants) | 92
  Cycle 2 Day 1: Post Dose | 36.0 (8.71)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 63
  Cycle 4 Day 1: Pre-dose | 5.41 (1.79)
  Cycle 4 Day 1: Post Dose: number analyzed (Participants) | 61
  Cycle 4 Day 1: Post Dose | 39.2 (7.30)

49. Secondary Outcome: Plasma Concentration of Polatuzumab Vedotin Analyte: Unconjugated MMAE
Description: PK of pola-related analytes unconjugated MMAE was measured. Cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts.
Time Frame: Cycle 1 Day 2: pre-dose and 30 min post dose, Cycle 1 Days 8 and 15; Cycles 2 and 4: pre-dose and 30 min post dose; unscheduled visits: pre-dose and 30 min post dose; study treatment completion (up to approximately 84 months)
Population: PK evaluable population included all the ITT participants Phase Ib and Phase II who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL | Arm A (Phase II Randomization): Pola+BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 36 | 36 | 18 | 18
ng/mL
  Cycle 1 Day 2: Pre-dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 35 | 36 | 17 | 17
  Cycle 1 Day 2: Pre-dose | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ.
  Cycle 1 Day 2: 30 min Post Dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 36 | 35 | 18 | 18
  Cycle 1 Day 2: 30 min Post Dose | 0.726 (297.5) | 0.234 (80.2) | 0.397 (67.7) | 0.327 (41.4) | 0.402 (80.2) | 0.315 (105.3) | 0.243 (101.8) | 0.456 (103.1)
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 6 | 6 | 6 | 0 | 0 | 0 | 0
  Cycle 1 Day 8 | 1.48 (100.8) | 1.84 (78.4) | 1.96 (51.5) | 2.34 (21.4) |  |  |  |
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 6 | 5 | 6 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 | 0.311 (93.8) | 0.531 (88.5) | 0.705 (60.0) | 0.688 (19.5) |  |  |  |
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 35 | 33 | 17 | 15
  Cycle 2 Day 1: Pre-dose | 0.0264 (70.8) | 0.158 (79.4) | 0.0512 (129.3) | 0.150 (44.4) | 0.0373 (81.5) | 0.159 (80.9) | 0.0451 (76.9) | 0.186 (86.8)
  Cycle 2 Day 1: 30 min Post Dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: 30 min Post Dose | 0.185 (54.2) | 0.263 (72.7) | 0.231 (53.5) | 0.345 (31.9) |  |  |  |
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 5 | 3 | 6 | 4 | 32 | 23 | 15 | 12
  Cycle 4 Day 1: Pre-dose | 0.0414 (102.9) | 0.133 (72.6) | 0.0511 (68.3) | 0.150 (44.3) | 0.0554 (77.3) | 0.158 (58.2) | 0.0481 (83.2) | 0.141 (102.3)
  Cycle 4 Day 1: 30 min Post Dose: number analyzed (Participants) | 4 | 3 | 6 | 4 | 29 | 23 | 15 | 12
  Cycle 4 Day 1: 30 min Post Dose | 0.234 (35.0) | 0.266 (27.0) | 0.167 (39.2) | 0.257 (32.3) | 0.198 (32.0) | 0.316 (38.9) | 0.195 (38.1) | 0.283 (56.9)
  Unscheduled Visit: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Unscheduled Visit |  |  |  |  |  |  | 0.738 (64.6) |
  Unscheduled Visit: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Unscheduled Visit: Pre-dose |  |  |  |  | 0.0180 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 0.0180 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  |
  Unscheduled Visit: 30 min Post Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Unscheduled Visit: 30 min Post Dose |  |  |  |  |  | 0.114 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  |
  Study Treatment Completion: number analyzed (Participants) | 0 | 0 | 1 | 0 | 28 | 27 | 13 | 8
  Study Treatment Completion |  |  | 0.0595 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 0.0506 (113.0) | 0.0749 (165.9) | 0.0682 (110.4) | 0.150 (179.4)

50. Secondary Outcome: Arm G+H (Phase II NF Cohorts): Plasma Concentration of Polatuzumab Vedotin Analyte: Unconjugated MMAE
Description: PK of one pola-related analytes: Unconjugated MMAE was measured. Cycle length is 21 days for DLBCL cohorts. As pre-specified in the protocol data is reported combined for arms G+H.
Time Frame: Cycle 1 Day 2: post dose; Cycle 1 and 3 Day 8 and 15; Cycle 2, 3 and 4 Day 1: pre-dose and post dose
Population: PK evaluable population included all the ITT participants in Arm G (Phase II NF Cohort) who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 103
ng/mL
  Cycle 1 Day 2: Post Dose | 0.590 (1.08)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 94
  Cycle 2 Day 1: Pre-dose | 0.229 (0.248)
  Cycle 2 Day 1: Post Dose: number analyzed (Participants) | 91
  Cycle 2 Day 1: Post Dose | 0.316 (0.213)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 61
  Cycle 4 Day 1: Pre-dose | 0.186 (0.118)
  Cycle 4 Day 1: Post Dose: number analyzed (Participants) | 60
  Cycle 4 Day 1: Post Dose | 0.256 (0.118)

51. Secondary Outcome: Plasma Concentration of Bendamustine
Description: Cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts. As pre specified in the protocol plasma concentration of bendamustine was not assessed in the Phase II NF Cohort (Arm G+H).
Time Frame: Cycle 1 Day 2: pre-dose, 5 min, 1 hour (h); 2h, 3h and 4h post dose
Population: as for outcome 47
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 37 | 39 | 35 | 33 | 18 | 19
ng/mL
  Cycle 1 Day 2: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 37 | 39 | 34 | 33 | 18 | 19
  Cycle 1 Day 2: Pre-dose |  |  |  |  | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ.
  Cycle 1 Day 2: 5 min Post Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 35 | 38 | 35 | 31 | 18 | 19
  Cycle 1 Day 2: 5 min Post Dose |  |  |  |  | 2130 (665.6) | 2810 (222.7) | 2740 (550.9) | 1700 (1865.5) | 3090 (68.3) | 3790 (119.4)
  Cycle 1 Day 2: 1h Post Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 35 | 39 | 34 | 31 | 17 | 18
  Cycle 1 Day 2: 1h Post Dose |  |  |  |  | 456 (167.8) | 353 (187.9) | 518 (154.2) | 451 (380.2) | 478 (111.4) | 639 (165.6)
  Cycle 1 Day 2: 2h Post Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 34 | 39 | 34 | 33 | 17 | 16
  Cycle 1 Day 2: 2h Post Dose |  |  |  |  | 84.4 (173.5) | 55.1 (236.5) | 93.8 (250.5) | 101 (375.8) | 62.8 (104.3) | 128 (196.7)
  Cycle 1 Day 2: 3h Post Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 33 | 38 | 34 | 32 | 17 | 15
  Cycle 1 Day 2: 3h Post Dose |  |  |  |  | 20.5 (220.1) | 12.7 (246.4) | 23.5 (461.0) | 21.5 (509.9) | 12.4 (132.0) | 28.2 (287.4)
  Cycle 1 Day 2: 4h Post Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 31 | 37 | 31 | 33 | 17 | 15
  Cycle 1 Day 2: 4h Post Dose |  |  |  |  | 7.60 (278.5) | 4.58 (268.4) | 8.11 (724.8) | 8.08 (615.9) | 3.30 (147.2) | 6.18 (131.0)

52. Secondary Outcome: Serum Concentration of Rituximab
Description: Cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts. As pre specified in the protocol serum concentration of rituximab was not assessed in the Phase II NF Cohort (Arm G+H).
Time Frame: Cycle 1 Days 1: pre-dose and 30 min post dose; Cycle 2 and 4 Day 1: pre-dose; unscheduled visits: pre-dose and 30 min post dose (up to approximately 84 months)
Population: PK evaluable population included all the ITT participants in Cohort 1a (Phase Ib) and Arms A-D (Phase II) who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL
Number analyzed (Participants) | 0 | 0 | 37 | 38 | 34 | 34
ng/mL
  Cycle 1 Days 1: Pre-dose |  |  | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ.
  Cycle 1 Days 1: 30 min Post Dose: number analyzed (Participants) | 0 | 0 | 32 | 38 | 34 | 33
  Cycle 1 Days 1: 30 min Post Dose |  |  | 182 (27.2) | 202 (24.5) | 188 (19.9) | 180 (18.0)
  Cycle 2 Days 1: Pre-dose: number analyzed (Participants) | 0 | 0 | 36 | 33 | 29 | 27
  Cycle 2 Days 1: Pre-dose |  |  | 22.8 (79.2) | 20.2 (145.9) | 34.9 (89.9) | 34.6 (69.7)
  Cycle 4 Days 1: Pre-dose: number analyzed (Participants) | 0 | 0 | 31 | 33 | 21 | 14
  Cycle 4 Days 1: Pre-dose |  |  | 65.1 (46.5) | 62.3 (42.7) | 74.7 (50.9) | 83.3 (49.1)
  Unscheduled: Pre-dose: number analyzed (Participants) | 0 | 0 | 2 | 0 | 1 | 1
  Unscheduled: Pre-dose |  |  | 30.6 (118.0) |  | 298 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 2.00 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated.
  Unscheduled: 30 min Post Dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Unscheduled: 30 min Post Dose |  |  |  |  |  | 165 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated.

53. Secondary Outcome: Serum Concentration of Obinutuzumab
Description: Cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts.
Time Frame: Cycles 1 and 4 Days 1: pre-dose and 30 min post dose; Cycle 2 Day1: pre-dose; Follow up visits on Day 1: Months 3, 6, 12, 18 and 24; unscheduled visits: pre-dose and 30 min post dose; study treatment completion (up to approximately 84 months)
Population: PK evaluable population included all the ITT participants who Cohort 1b (Phase 1b) and Arms E and F (Phase II) received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: g/mL
Arm/Group | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL
Number analyzed (Participants) | 6 | 6 | 19 | 19
g/mL
  Cycle 1 Day 1: Pre-dose: number analyzed (Participants) | 6 | 5 | 19 | 19
  Cycle 1 Day 1: Pre-dose | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ.
  Cycle 1 Day 1: 30 min Post Dose: number analyzed (Participants) | 0 | 0 | 14 | 13
  Cycle 1 Day 1: 30 min Post Dose |  |  | 341 (22.1) | 221 (105.5)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 6 | 6 | 18 | 17
  Cycle 2 Day 1: Pre-dose | 283 (38.4) | 412 (40.8) | 301 (39.3) | 349 (58.0)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 6 | 4 | 17 | 12
  Cycle 4 Day 1: Pre-dose | 293 (53.8) | 359 (28.9) | 291 (37.9) | 290 (36.4)
  Cycle 4 Day 1: 30 min Post Dose: number analyzed (Participants) | 0 | 0 | 16 | 12
  Cycle 4 Day 1: 30 min Post Dose |  |  | 701 (27.4) | 642 (29.5)
  Follow up on Month 3, Day 1: number analyzed (Participants) | 5 | 2 | 16 | 8
  Follow up on Month 3, Day 1 | 67.7 (47.8) | 28.8 (17.0) | 38.5 (167.8) | 55.1 (119.9)
  Follow up on Month 6, Day 1: number analyzed (Participants) | 5 | 2 | 10 | 7
  Follow up on Month 6, Day 1 | 11.5 (56.6) | 5.38 (12.4) | 7.64 (412.2) | 15.8 (137.6)
  Follow up on Month 12, Day 1: number analyzed (Participants) | 4 | 3 | 6 | 2
  Follow up on Month 12, Day 1 | 0.237 (717.6) | 0.389 (119.3) | 0.162 (569.7) | 0.732 (18.7)
  Follow up on Month 18, Day 1: number analyzed (Participants) | 2 | 2 | 7 | 3
  Follow up on Month 18, Day 1 | 0.00978 (1188.5) | 0.0107 (170.5) | 0.00842 (347.4) | 0.0460 (86.9)
  Follow up on Month 24, Day 1: number analyzed (Participants) | 1 | 1 | 0 | 1
  Follow up on Month 24, Day 1 | 0.00203 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 0.00203 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 0.00203 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated.
  Unscheduled: number analyzed (Participants) | 0 | 1 | 1 | 0
  Unscheduled |  | 3.09 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 20.8 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |
  Unscheduled Visit: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Unscheduled Visit: Pre-dose |  |  |  | 0.0626 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated.
  Unscheduled Visit: 30 min Post Dose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Unscheduled Visit: 30 min Post Dose |  |  |  | 349 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated.
  Study Treatment Completion Visit: number analyzed (Participants) | 1 | 0 | 14 | 8
  Study Treatment Completion Visit | 367 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 242 (52.7) | 232 (46.2)

54. Secondary Outcome: Phase Ib: Cmax of Polatuzumab Vedotin, Bendamustine, and Rituximab in Cohort 1a
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Cycles 1, 2 and 4 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Cohort 1a (Phase Ib) who received at least one study treatment and who provided suitable PK samples. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema Cmax was not evaluated for Bendamustine and Rituximab.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL
Number analyzed (Participants) | 6 | 6
ng/mL
  acMMAE: Cycle 1 | 676 (176) | 634 (158)
  acMMAE: Cycle 2 | 697 (129) | 694 (138)
  acMMAE: Cycle 4: number analyzed (Participants) | 5 | 3
  acMMAE: Cycle 4 | 763 (159) | 759 (107)
  Total Ab: Cycle 1 | 34.3 (8.57) | 37.6 (9.42)
  Total Ab: Cycle 2 | 36.6 (8.00) | 40.6 (9.46)
  Total Ab: Cycle 4: number analyzed (Participants) | 5 | 3
  Total Ab: Cycle 4 | 41.3 (9.98) | 44.8 (5.06)
  Unconjugated MMAE: Cycle 1 | 3.31 (4.00) | 2.21 (1.34)
  Unconjugated MMAE: Cycle 2: number analyzed (Participants) | 0 | 0
  Unconjugated MMAE: Cycle 4: number analyzed (Participants) | 0 | 0
  Bendamustine: Cycle 1: number analyzed (Participants) | 0 | 0
  Bendamustine: Cycle 2: number analyzed (Participants) | 0 | 0
  Bendamustine: Cycle 4: number analyzed (Participants) | 0 | 0
  Rituximab: Cycle 1: number analyzed (Participants) | 0 | 0
  Rituximab: Cycle 2: number analyzed (Participants) | 0 | 0
  Rituximab: Cycle 4: number analyzed (Participants) | 0 | 0

55. Secondary Outcome: Phase Ib: Cmax of Polatuzumab Vedotin, Bendamustine, and Obinutuzumab in Cohort 1b
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Cycles 1, 2 and 4 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants Cohort 1b (Phase Ib) who received at least one study treatment and who provided suitable PK samples. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema Cmax was not evaluated for Bendamustine and Obinutuzumab.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL
Number analyzed (Participants) | 6 | 6
ng/mL
  acMMAE: Cycle 1 | 738 (165) | 725 (104)
  acMMAE: Cycle 2 | 816 (168) | 841 (115)
  acMMAE: Cycle 4: number analyzed (Participants) | 6 | 4
  acMMAE: Cycle 4 | 749 (158) | 721 (97.7)
  Total Ab: Cycle 1 | 38.7 (9.84) | 34.9 (7.52)
  Total Ab: Cycle 2 | 45.0 (12.1) | 43.1 (9.52)
  Total Ab: Cycle 4: number analyzed (Participants) | 6 | 4
  Total Ab: Cycle 4 | 44.2 (11.2) | 48.2 (12.5)
  Unconjugated MMAE: Cycle 1 | 2.17 (1.08) | 2.39 (0.492)
  Unconjugated MMAE: Cycle 2: number analyzed (Participants) | 0 | 0
  Unconjugated MMAE: Cycle 4: number analyzed (Participants) | 0 | 0
  Bendamustine: Cycle 1: number analyzed (Participants) | 0 | 0
  Bendamustine: Cycle 2: number analyzed (Participants) | 0 | 0
  Bendamustine: Cycle 4: number analyzed (Participants) | 0 | 0
  Rituximab: Cycle 1: number analyzed (Participants) | 0 | 0
  Rituximab: Cycle 2: number analyzed (Participants) | 0 | 0
  Rituximab: Cycle 4: number analyzed (Participants) | 0 | 0

56. Secondary Outcome: Phase II: Cmax of Polatuzumab Vedotin, Bendamustine, and Rituximab in Arms A and C
Description: PK of three pola-related analytes: acMMAE, total antibody and unconjugated MMAE were measured.
Time Frame: Cycle 1; Cycle 4 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Arms A and C who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL
Number analyzed (Participants) | 36 | 35
ng/mL
  acMMAE: Cycle 1 | 622 (194) | 661 (149)
  acMMAE: Cycle 4: number analyzed (Participants) | 29 | 23
  acMMAE: Cycle 4 | 703 (150) | 659 (135)
  Total Ab: Cycle 1 | 36.7 (9.54) | 35.7 (8.50)
  Total Ab: Cycle 4: number analyzed (Participants) | 31 | 23
  Total Ab: Cycle 4 | 46.1 (11.4) | 41.4 (8.29)
  Unconjugated MMAE: Cycle 1: number analyzed (Participants) | 0 | 0
  Unconjugated MMAE: Cycle 4: number analyzed (Participants) | 0 | 0
  Bendamustine: Cycle 1: number analyzed (Participants) | 34 | 33
  Bendamustine: Cycle 1 | 3.57 (2.06) | 4.23 (2.26)
  Bendamustine: Cycle 4: number analyzed (Participants) | 0 | 0
  Rituximab: Cycle 1: number analyzed (Participants) | 32 | 34
  Rituximab: Cycle 1 | 188 (49.2) | 191 (35.9)
  Rituximab: Cycle 4: number analyzed (Participants) | 0 | 0

57. Secondary Outcome: Phase II: Cmax of Bendamustine and Rituximab in Arms B and D
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Arms B and D who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Arm B (Phase II Randomization): BR in FL | Arm D (Phase II Randomization): BR in DLBCL
Number analyzed (Participants) | 38 | 33
ug/mL
  Bendamustine: number analyzed (Participants) | 34 | 30
  Bendamustine | 3.21 (2.09) | 3.85 (2.91)
  Rituximab | 207 (50.1) | 183 (33.6)

58. Secondary Outcome: Phase II: Cmax of Polatuzumab Vedotin, Obinutuzumab and Bendamustine in Arms E and F
Description: PK of three pola-related analytes: acMMAE, unconjugated MMAE and total antibody were measured.
Time Frame: Cycle 1; Cycle 4 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Arms E and F who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL
Number analyzed (Participants) | 18 | 19
ug/mL
  acMMAE: Cycle 1 | 692 (230) | 703 (211)
  acMMAE: Cycle 4: number analyzed (Participants) | 17 | 12
  acMMAE: Cycle 4 | 845 (165) | 713 (70.6)
  Total Ab: Cycle 1 | 33.3 (8.04) | 39.0 (7.63)
  Total Ab: Cycle 4: number analyzed (Participants) | 17 | 12
  Total Ab: Cycle 4 | 56.1 (11.2) | 37.8 (4.51)
  Unconjugated MMAE: Cycle 1: number analyzed (Participants) | 0 | 0
  Unconjugated MMAE: Cycle 4: number analyzed (Participants) | 0 | 0
  Bendamustine: Cycle 1: number analyzed (Participants) | 16 | 19
  Bendamustine: Cycle 1 | 3.30 (1.58) | 5.47 (4.30)
  Bendamustine: Cycle 4: number analyzed (Participants) | 0 | 0
  Obinutuzumab: Cycle 1: number analyzed (Participants) | 14 | 13
  Obinutuzumab: Cycle 1 | 349 (72.8) | 274 (118)
  Obinutuzumab: Cycle 4: number analyzed (Participants) | 16 | 12
  Obinutuzumab: Cycle 4 | 727 (217) | 666 (190)

59. Secondary Outcome: Arm H (Phase II NF Cohort): Cmax of Polatuzumab Vedotin (Lyophilized)
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: as for outcome 9
Population: as for outcome 11
Arm/Group | Arm H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 0

60. Secondary Outcome: Phase Ib: AUC From Time Zero to Infinity (AUCinf) of Polatuzumab Vedotin, Bendamustine, and Rituximab in Cohort 1a
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured. The unit of measure for AUC is day*micrograms per milliliter [day*ug/mL]).
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Cohort 1a (Phase Ib) who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema AUC was not evaluated for bendamustine and rituximab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL
Number analyzed (Participants) | 4 | 6
day*ug/mL
  acMMAE | 2830 (12.1) | 2110 (28.4)
  Total Ab | 298 (4.9) | 214 (35.9)
  Unconjugated MMAE: number analyzed (Participants) | 0 | 0
  Bendamustine: number analyzed (Participants) | 0 | 0
  Rituximab: number analyzed (Participants) | 0 | 0

61. Secondary Outcome: Phase Ib: AUCinf of Polatuzumab Vedotin, Bendamustine, and Obinutuzumab in Cohort 1b
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Cohort 1b (Phase Ib) who received at least one study treatment and who provided suitable PK samples. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema AUC was not evaluated for bendamustine and obinutuzumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL
Number analyzed (Participants) | 6 | 6
day*ug/mL
  acMMAE: number analyzed (Participants) | 5 | 6
  acMMAE | 2600 (34.4) | 2650 (16.4)
  Total Ab | 267 (30.2) | 252 (21.6)
  Unconjugated MMAE: number analyzed (Participants) | 0 | 0
  Bendamustine: number analyzed (Participants) | 0 | 0
  Obinutuzumab: number analyzed (Participants) | 0 | 0

62. Secondary Outcome: Phase II: AUCinf of Polatuzumab Vedotin, Bendamustine, and Rituximab in Arms A and C
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Arms A and C who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema AUC was not evaluated for pola and rituximab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL
Number analyzed (Participants) | 31 | 30
h*ug/mL
  acMMAE: number analyzed (Participants) | 0 | 0
  Total Ab: number analyzed (Participants) | 0 | 0
  Unconjugated MMAE: number analyzed (Participants) | 0 | 0
  Bendamustine | 3.29 (73.3) | 3.62 (78.5)
  Rituximab: number analyzed (Participants) | 0 | 0

63. Secondary Outcome: Phase II: AUCinf of Bendamustine and Rituximab in Arms B and D
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Arms B and D who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema AUC was not evaluated for rituximab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Arm B (Phase II Randomization): BR in FL | Arm D (Phase II Randomization): BR in DLBCL
Number analyzed (Participants) | 33 | 29
h*ug/mL
  Bendamustine | 2.86 (67.3) | 3.43 (97.4)
  Rituximab: number analyzed (Participants) | 0 | 0

64. Secondary Outcome: Phase II: AUCinf of Polatuzumab Vedotin, Bendamustine, and Obinutuzumab in Arms E and F
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Arms E and F who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema AUC was not evaluated for pola and obinutuzumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL
Number analyzed (Participants) | 15 | 14
h*ug/mL
  acMMAE: number analyzed (Participants) | 0 | 0
  Total Ab: number analyzed (Participants) | 0 | 0
  Unconjugated MMAE: number analyzed (Participants) | 0 | 0
  Bendamustine | 2.88 (28.9) | 4.10 (67.4)
  Obinutuzumab: number analyzed (Participants) | 0 | 0

65. Secondary Outcome: Arm H (Phase II NF Cohort): AUC of Polatuzumab Vedotin (Lyophilized)
Description: PK of three pola-related analytes: antibody acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Days 2, 8 and 15 of Cycle 1, Day 1 of Cycle 2 and 4, (each cycle is 21 days DLBCL cohorts) up to approximately 9 weeks
Population: as for outcome 11
Arm/Group | Arm H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 0

66. Secondary Outcome: Phase Ib: CL of Polatuzumab Vedotin, Bendamustine, and Rituximab in Cohort 1a
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Cohort 1a (Phase Ib) who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema CL was not evaluated for bendamustine and rituximab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day/kg
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL
Number analyzed (Participants) | 4 | 6
mL/day/kg
  acMMAE | 11.3 (12.9) | 15.2 (27.9)
  Total Ab | 6.05 (4.7) | 8.48 (35.2)
  Unconjugated MMAE: number analyzed (Participants) | 0 | 0
  Bendamustine: number analyzed (Participants) | 0 | 0
  Rituximab: number analyzed (Participants) | 0 | 0

67. Secondary Outcome: Phase Ib: CL of Polatuzumab Vedotin, Bendamustine, and Obinutuzumab in Cohort 1b
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Cohort 1b (Phase Ib) who received at least one study treatment and who provided suitable PK samples. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema CL was not evaluated for bendamustine and obinutuzumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day/kg
Arm/Group | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL
Number analyzed (Participants) | 6 | 6
mL/day/kg
  acMMAE: number analyzed (Participants) | 5 | 6
  acMMAE | 12.3 (34.9) | 12.1 (17.0)
  Total Ab | 6.76 (30.6) | 7.17 (22.2)
  Unconjugated MMAE: number analyzed (Participants) | 0 | 0
  Bendamustine: number analyzed (Participants) | 0 | 0
  Obinutuzumab: number analyzed (Participants) | 0 | 0

68. Secondary Outcome: Phase II: CL of Polatuzumab Vedotin, Bendamustine and Rituximab in Arms A and C
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Arms A and B who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema CL was not evaluated for pola and rituximab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/h)
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL
Number analyzed (Participants) | 30 | 29
Liters per hour (L/h)
  acMMAE: number analyzed (Participants) | 0 | 0
  Total Ab: number analyzed (Participants) | 0 | 0
  Unconjugated MMAE: number analyzed (Participants) | 0 | 0
  Bendamustine | 47.9 (60.8) | 42.6 (66.4)
  Rituximab: number analyzed (Participants) | 0 | 0

69. Secondary Outcome: Phase II: CL of Bendamustine and Rituximab in Arms B and D
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Arms B and D who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema CL was not evaluated for rituximab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Arm B (Phase II Randomization): BR in FL | Arm D (Phase II Randomization): BR in DLBCL
Number analyzed (Participants) | 32 | 29
L/h
  Bendamustine | 54.4 (60.9) | 46.4 (93.9)
  Rituximab: number analyzed (Participants) | 0 | 0

70. Secondary Outcome: Phase II: CL of Polatuzumab Vedotin, Bendamustine and Obinutuzumab in Arms E and F
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: as for outcome 64
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL
Number analyzed (Participants) | 15 | 14
L/h
  acMMAE: number analyzed (Participants) | 0 | 0
  Total Ab: number analyzed (Participants) | 0 | 0
  Uncojugated MMAE: number analyzed (Participants) | 0 | 0
  Bendamustine | 61.3 (33.4) | 39.9 (76.1)
  Obinutuzumab: number analyzed (Participants) | 0 | 0

71. Secondary Outcome: Arm H (Phase II NF Cohort): CL of Polatuzumab Vedotin (Lyophilized)
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: as for outcome 10
Population: as for outcome 11
Arm/Group | Arm H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 0

72. Secondary Outcome: Phase Ib: Vss of Polatuzumab Vedotin, Bendamustine, and Obinutuzumab in Cohort 1a
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Cohort 1a (Phase Ib) who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema Vss was not evaluated for bendamustine and rituximab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL
Number analyzed (Participants) | 4 | 6
mL/kg
  acMMAE | 73.0 (22.3) | 82.7 (33.2)
  Total Ab | 82.3 (9.1) | 76.6 (25.7)
  Unconjugated MMAE: number analyzed (Participants) | 0 | 0
  Bendamustine: number analyzed (Participants) | 0 | 0
  Rituximab: number analyzed (Participants) | 0 | 0

73. Secondary Outcome: Phase Ib: Vss of Polatuzumab Vedotin, Bendamustine, and Obinutuzumab in Cohort 1b
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Cohort 1b (Phase Ib) who received at least one study treatment and who provided suitable PK samples. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema Vss was not evaluated for bendamustine and obinutuzumab.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL
Number analyzed (Participants) | 6 | 6
mL/kg
  acMMAE: number analyzed (Participants) | 5 | 6
  acMMAE | 77.2 (38.8) | 64.7 (23.0)
  Total Ab | 87.5 (38.5) | 87.9 (24.7)
  Unconjugated MMAE: number analyzed (Participants) | 0 | 0
  Bendamustine: number analyzed (Participants) | 0 | 0
  Obinutuzumab: number analyzed (Participants) | 0 | 0

74. Secondary Outcome: Phase II: Vss of Polatuzumab Vedotin, Bendamustine and Rituximab in Arms A and C
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Arms A and C who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema Vss was not evaluated for pola and rituximab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL
Number analyzed (Participants) | 29 | 29
L
  acMMAE: number analyzed (Participants) | 0 | 0
  Total Ab: number analyzed (Participants) | 0 | 0
  Unconjugated MMAE: number analyzed (Participants) | 0 | 0
  Bendamustine | 36.5 (86.4) | 34.3 (57.7)
  Rituximab: number analyzed (Participants) | 0 | 0

75. Secondary Outcome: Phase II: Vss of Bendamustine and Rituximab in Arms B and D
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Arms B and D who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema Vss was not evaluated for rituximab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Arm B (Phase II Randomization): BR in FL | Arm D (Phase II Randomization): BR in DLBCL
Number analyzed (Participants) | 31 | 24
L
  Bendamustine | 44.9 (69.6) | 33.2 (62.9)
  Rituximab: number analyzed (Participants) | 0 | 0

76. Secondary Outcome: Phase II: Vss of Polatuzumab Vedotin, Bendamustine and Obinutuzumab in Arms E and F
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: Cycle 1 Day 2 (cycle length is 21 days for DLBCL cohorts and 28 days for FL cohorts)
Population: PK evaluable population included all the ITT participants in Arms E and F who received at least one study treatment and who provided suitable PK samples. 'Overall Number Analyzed' are the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoints. Due to the sparse sample collection schema Vss was not evaluated for pola and obinutuzumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL
Number analyzed (Participants) | 14 | 12
L
  acMMAE: number analyzed (Participants) | 0 | 0
  Total Ab: number analyzed (Participants) | 0 | 0
  Unconjugated MMAE: number analyzed (Participants) | 0 | 0
  Bendamustine | 51.2 (33.6) | 31.5 (68.1)
  Obinutuzumab: number analyzed (Participants) | 0 | 0

77. Secondary Outcome: Arm H (Phase II NF Cohort): Vss of Polatuzumab Vedotin (Lyophilized)
Description: PK of three pola-related analytes: acMMAE, total antibody, and unconjugated MMAE were measured.
Time Frame: as for outcome 11
Population: as for outcome 11
Arm/Group | Arm H (Phase II NF Cohort): Pola+BR in DLBCL
Number analyzed (Participants) | 0

78. Secondary Outcome: Symptom Severity and Interference According to Therapy-Induced Neuropathy Assessment Score (TINAS) in Arms A-F
Description: The TINAS is an 11-item questionnaire that assesses the severity of neuropathy-related symptoms in the last 24 hours. The 11 items assessed were: hot/burning sensations in hands/feet, sensations pins and needles arms/legs, numbness or tingling in hands/feet, sensations of electric shock, pain when touching cold things, cramps in hands/feet, discomfort when touching things, discomfort skin contact with something, trouble grasping small objects, trouble walking loss feeling legs/feet, difficulty balance loss feeling leg/feet. Each item was scored on a 0-10 scale, with 0 being the symptom is not present, and 10 being the symptom is as bad as the participant can imagine. Higher scores indicate more severe disease. Scores were averaged at each week.
Time Frame: Every week during treatment (up to 24 weeks) and for the first 2 months after treatment, thereafter every month for 10 months or until withdrawal (up to 18 months overall)
Population: ITT population included all randomized participants in Arms A-F (Phase II) irrespective of whether or not they received the study treatment. 'Overall Number Analysed' =number of participants with data available for analysis. 'Number of Participants Analyzed'=number of participants evaluable for this outcome measure. Participants from Arm F did not answer a sufficient number of questions at both baseline and end of treatment visit therefore the average score could not be calculated.
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL
Number analyzed (Participants) | 15 | 14 | 11 | 12 | 5 | 0
Points on scale
  Baseline | 0.2 (0.3) | 0.5 (1.1) | 0.4 (0.6) | 0.6 (0.7) | 0.8 (1.6) |
  Week 1: number analyzed (Participants) | 2 | 0 | 0 | 0 | 1 | 0
  Week 1 | 0.3 (0.4) |  |  |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 2: number analyzed (Participants) | 13 | 13 | 10 | 11 | 3 | 0
  Week 2 | 0.3 (0.4) | 0.5 (1.3) | 0.3 (0.4) | 1.0 (1.1) | 0.2 (0.2) |
  Week 3: number analyzed (Participants) | 15 | 13 | 7 | 10 | 4 | 0
  Week 3 | 0.2 (0.5) | 0.7 (1.5) | 0.1 (0.1) | 0.9 (0.1) | 0.0 (0.1) |
  Week 4: number analyzed (Participants) | 12 | 13 | 8 | 9 | 5 | 0
  Week 4 | 0.1 (0.2) | 0.8 (1.8) | 0.3 (0.3) | 0.7 (0.8) | 0.2 (0.4) |
  Week 5: number analyzed (Participants) | 14 | 13 | 8 | 8 | 4 | 0
  Week 5 | 0.2 (0.3) | 0.6 (1.4) | 0.3 (0.5) | 0.6 (0.6) | 0.1 (0.2) |
  Week 6: number analyzed (Participants) | 12 | 13 | 8 | 8 | 4 | 0
  Week 6 | 0.2 (0.4) | 0.8 (1.8) | 0.3 (0.5) | 0.7 (1.0) | 0.1 (0.3) |
  Week 7: number analyzed (Participants) | 11 | 11 | 8 | 8 | 4 | 0
  Week 7 | 0.3 (0.4) | 0.9 (1.9) | 0.2 (0.3) | 0.4 (0.6) | 0.0 (0.1) |
  Week 8: number analyzed (Participants) | 13 | 12 | 7 | 7 | 4 | 0
  Week 8 | 0.3 (0.4) | 0.8 (1.8) | 0.2 (0.5) | 0.6 (0.9) | 0.2 (0.4) |
  Week 9: number analyzed (Participants) | 14 | 14 | 7 | 6 | 5 | 0
  Week 9 | 0.4 (0.9) | 0.5 (0.9) | 0.2 (0.3) | 0.5 (0.7) | 0.1 (0.3) |
  Week 10: number analyzed (Participants) | 12 | 13 | 7 | 6 | 3 | 0
  Week 10 | 0.5 (0.9) | 0.4 (0.8) | 0.1 (0.1) | 0.2 (0.4) | 0.1 (0.2) |
  Week 11: number analyzed (Participants) | 14 | 13 | 8 | 6 | 5 | 0
  Week 11 | 0.5 (1.0) | 0.5 (0.9) | 0.2 (0.2) | 0.4 (0.6) | 0.1 (0.1) |
  Week 12: number analyzed (Participants) | 13 | 12 | 6 | 5 | 3 | 0
  Week 12 | 0.5 (1.4) | 0.9 (2.0) | 0.3 (0.4) | 0.3 (0.6) | 0.2 (0.2) |
  Week 13: number analyzed (Participants) | 12 | 14 | 7 | 5 | 4 | 0
  Week 13 | 0.7 (1.2) | 0.6 (1.6) | 0.3 (0.4) | 0.2 (0.4) | 0.3 (0.4) |
  Week 14: number analyzed (Participants) | 12 | 11 | 7 | 5 | 5 | 0
  Week 14 | 0.6 (1.2) | 0.7 (1.8) | 0.3 (0.3) | 0.4 (0.6) | 0.2 (0.4) |
  Week 15: number analyzed (Participants) | 11 | 12 | 7 | 5 | 3 | 0
  Week 15 | 0.2 (0.3) | 0.7 (1.7) | 0.4 (0.5) | 0.4 (0.4) | 0.9 (1.6) |
  Week 16: number analyzed (Participants) | 11 | 11 | 5 | 5 | 5 | 0
  Week 16 | 0.4 (0.5) | 0.8 (1.8) | 0.4 (0.4) | 0.4 (0.5) | 0.3 (0.7) |
  Week 17: number analyzed (Participants) | 11 | 11 | 6 | 5 | 4 | 0
  Week 17 | 0.2 (0.3) | 0.8 (1.8) | 0.5 (0.7) | 0.4 (0.6) | 0.3 (0.5) |
  Week 18: number analyzed (Participants) | 10 | 11 | 6 | 2 | 4 | 0
  Week 18 | 0.2 (0.3) | 0.7 (1.8) | 0.3 (0.4) | 0.1 (0.1) | 0.3 (0.5) |
  Week 19: number analyzed (Participants) | 12 | 9 | 6 | 4 | 4 | 0
  Week 19 | 0.2 (0.3) | 0.8 (2.0) | 0.4 (0.7) | 0.5 (0.8) | 0.3 (0.5) |
  Week 20: number analyzed (Participants) | 11 | 9 | 5 | 3 | 4 | 0
  Week 20 | 0.0 (0.2) | 0.8 (1.9) | 0.6 (0.8) | 0.1 (0.1) | 0.3 (0.4) |
  Week 21: number analyzed (Participants) | 7 | 10 | 5 | 3 | 4 | 0
  Week 21 | 0.3 (0.3) | 0.9 (1.9) | 0.5 (0.5) | 0.1 (0.1) | 0.3 (0.3) |
  Week 22: number analyzed (Participants) | 9 | 9 | 3 | 1 | 3 | 0
  Week 22 | 0.2 (0.2) | 0.8 (2.0) | 0.9 (1.5) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.5 (0.6) |
  Week 23: number analyzed (Participants) | 7 | 9 | 7 | 1 | 3 | 0
  Week 23 | 0.2 (0.3) | 0.8 (2.2) | 0.6 (0.7) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.5 (0.6) |
  Week 24: number analyzed (Participants) | 7 | 8 | 7 | 2 | 4 | 0
  Week 24 | 0.4 (0.6) | 1.0 (2.3) | 0.5 (0.7) | 0.0 (0.1) | 0.3 (0.3) |
  Week 25: number analyzed (Participants) | 8 | 7 | 6 | 1 | 2 | 0
  Week 25 | 0.2 (0.2) | 0.2 (0.2) | 0.3 (0.4) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.1 (0.1) |
  Week 26: number analyzed (Participants) | 5 | 2 | 7 | 1 | 0 | 0
  Week 26 | 0.6 (0.8) | 3.3 (4.4) | 0.4 (0.6) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  |
  Week 27: number analyzed (Participants) | 7 | 7 | 6 | 2 | 3 | 0
  Week 27 | 0.3 (0.3) | 1.1 (2.5) | 0.5 (0.6) | 0.1 (0.1) | 0.4 (0.4) |
  Week 28: number analyzed (Participants) | 8 | 6 | 7 | 1 | 2 | 0
  Week 28 | 0.5 (0.6) | 1.2 (2.6) | 0.5 (0.7) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.1 (0.2) |
  Week 29: number analyzed (Participants) | 8 | 7 | 7 | 1 | 3 | 0
  Week 29 | 0.2 (0.2) | 0.8 (2.1) | 0.7 (0.7) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.1 (0.2) |
  Week 30: number analyzed (Participants) | 6 | 8 | 4 | 1 | 2 | 0
  Week 30 | 0.7 (1.1) | 0.7 (1.9) | 0.8 (0.8) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.1 (0.1) |
  Week 31: number analyzed (Participants) | 7 | 4 | 3 | 1 | 3 | 0
  Week 31 | 0.3 (0.3) | 0.0 (0.1) | 1.3 (0.9) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.1 (0.1) |
  Week 32: number analyzed (Participants) | 5 | 6 | 4 | 0 | 2 | 0
  Week 32 | 0.4 (0.4) | 0.1 (0.1) | 1.0 (0.9) |  | 0.2 (0.3) |
  Week 33: number analyzed (Participants) | 4 | 6 | 4 | 0 | 3 | 0
  Week 33 | 0.3 (0.3) | 0.1 (0.2) | 1.0 (1.0) |  | 0.2 (0.2) |
  Week 34: number analyzed (Participants) | 6 | 4 | 3 | 0 | 2 | 0
  Week 34 | 0.2 (0.2) | 1.3 (2.4) | 0.8 (0.5) |  | 0.2 (0.3) |
  Week 35: number analyzed (Participants) | 4 | 1 | 3 | 2 | 1 | 0
  Week 35 | 0.3 (0.3) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 1.2 (0.7) | 0.6 (0.9) | 0.4 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 36: number analyzed (Participants) | 3 | 2 | 3 | 0 | 2 | 0
  Week 36 | 0.5 (0.3) | 0.2 (0.3) | 1.2 (0.6) |  | 0.1 (0.2) |
  Week 37: number analyzed (Participants) | 3 | 5 | 4 | 0 | 2 | 0
  Week 37 | 0.4 (0.4) | 0.1 (0.1) | 1.1 (0.8) |  | 0.2 (0.3) |
  Week 38: number analyzed (Participants) | 3 | 1 | 2 | 0 | 1 | 0
  Week 38 | 0.4 (0.4) | 0.1 (NA) — SD is not evaluable when only one participant is analyzed | 1.5 (0.4) |  | 0.3 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 39: number analyzed (Participants) | 5 | 1 | 2 | 1 | 1 | 0
  Week 39 | 0.7 (0.9) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 1.5 (0.5) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.3 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 40: number analyzed (Participants) | 3 | 1 | 3 | 0 | 2 | 0
  Week 40 | 0.5 (0.4) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.9 (0.4) |  | 0.1 (0.2) |
  Week 41: number analyzed (Participants) | 2 | 7 | 4 | 0 | 2 | 0
  Week 41 | 0.6 (0.6) | 0.7 (1.6) | 1.4 (1.2) |  | 0.3 (0.4) |
  Week 42: number analyzed (Participants) | 3 | 1 | 1 | 0 | 1 | 0
  Week 42 | 0.5 (0.5) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.3 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.5 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 43: number analyzed (Participants) | 4 | 1 | 1 | 1 | 1 | 0
  Week 43 | 0.3 (0.4) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.6 (NA) — SD is not evaluable when only one participant is analyzed | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.4 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 44: number analyzed (Participants) | 1 | 1 | 2 | 0 | 1 | 0
  Week 44 | 1.6 (NA) — SD is not evaluable when only one participant is analyzed | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.2 (0.3) |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 45: number analyzed (Participants) | 3 | 7 | 2 | 0 | 2 | 0
  Week 45 | 0.8 (0.7) | 0.1 (0.2) | 1.0 (1.2) |  | 0.3 (0.4) |
  Week 46: number analyzed (Participants) | 2 | 1 | 1 | 0 | 1 | 0
  Week 46 | 1.1 (0.7) | 0.1 (NA) — SD is not evaluable when only one participant is analyzed | 0.2 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.5 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 47: number analyzed (Participants) | 4 | 1 | 1 | 0 | 1 | 0
  Week 47 | 0.4 (0.6) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.1 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.8 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 48: number analyzed (Participants) | 0 | 2 | 3 | 0 | 1 | 0
  Week 48 |  | 0.8 (0.9) | 0.2 (0.2) |  | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 49: number analyzed (Participants) | 2 | 7 | 2 | 0 | 2 | 0
  Week 49 | 0.6 (0.6) | 0.0 (0.0) | 1.1 (1.4) |  | 0.3 (0.4) |
  Week 50: number analyzed (Participants) | 2 | 1 | 1 | 0 | 1 | 0
  Week 50 | 1.0 (0.2) | 0.1 (NA) — SD is not evaluable when only one participant is analyzed | 0.2 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.5 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 51: number analyzed (Participants) | 2 | 1 | 1 | 0 | 1 | 0
  Week 51 | 0.1 (0.2) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.2 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.5 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 52: number analyzed (Participants) | 1 | 2 | 1 | 0 | 1 | 0
  Week 52 | 0.4 (NA) — SD is not evaluable when only one participant is analyzed | 0.4 (0.5) | 0.2 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.5 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 53: number analyzed (Participants) | 1 | 5 | 1 | 0 | 2 | 0
  Week 53 | 0.2 (NA) — SD is not evaluable when only one participant is analyzed | 0.7 (1.5) | 0.2 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.2 (0.3) |
  Week 54: number analyzed (Participants) | 2 | 1 | 1 | 0 | 1 | 0
  Week 54 | 0.8 (0.6) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.2 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.5 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 55: number analyzed (Participants) | 2 | 1 | 1 | 0 | 1 | 0
  Week 55 | 0.3 (0.5) | 0.2 (NA) — SD is not evaluable when only one participant is analyzed | 0.2 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.5 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 56: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  Week 56 | 0.6 (0.3) | 0.2 (NA) — SD is not evaluable when only one participant is analyzed | 0.0 (0.1) |  |  |
  Week 57: number analyzed (Participants) | 1 | 6 | 2 | 0 | 2 | 0
  Week 57 | 0.3 (NA) — SD is not evaluable when only one participant is analyzed | 0.0 (0.0) | 1.5 (2.1) |  | 0.2 (0.3) |
  Week 58: number analyzed (Participants) | 4 | 0 | 1 | 0 | 1 | 0
  Week 58 | 0.7 (0.6) |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 59: number analyzed (Participants) | 2 | 1 | 1 | 0 | 1 | 0
  Week 59 | 0.0 (0.1) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 60: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0
  Week 60 | 0.4 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  |  |
  Week 61: number analyzed (Participants) | 3 | 6 | 2 | 0 | 2 | 0
  Week 61 | 0.4 (0.3) | 0.3 (0.5) | 1.5 (2.1) |  | 0.3 (0.5) |
  Week 62: number analyzed (Participants) | 2 | 0 | 1 | 0 | 1 | 0
  Week 62 | 0.7 (1.0) |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 63: number analyzed (Participants) | 3 | 1 | 1 | 0 | 1 | 0
  Week 63 | 0.4 (0.7) | 0.0 (NA) — SD is not evaluable when only one participant is analyzed | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.8 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 64: number analyzed (Participants) | 1 | 1 | 2 | 0 | 1 | 0
  Week 64 | 0.4 (NA) — SD is not evaluable when only one participant is analyzed | 1.1 (NA) — SD is not evaluable when only one participant is analyzed | 0.1 (0.2) |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 65: number analyzed (Participants) | 2 | 4 | 3 | 0 | 1 | 0
  Week 65 | 0.2 (0.0) | 0.0 (0.0) | 0.8 (1.3) |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 66: number analyzed (Participants) | 3 | 0 | 1 | 0 | 1 | 0
  Week 66 | 0.6 (0.7) |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.8 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 67: number analyzed (Participants) | 2 | 0 | 1 | 0 | 1 | 0
  Week 67 | 0.2 (0.3) |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.9 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 68: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 68 |  |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 1.2 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 69: number analyzed (Participants) | 1 | 5 | 2 | 0 | 1 | 0
  Week 69 | 0.2 (NA) — SD is not evaluable when only one participant is analyzed | 0.3 (0.5) | 1.5 (2.1) |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 70: number analyzed (Participants) | 2 | 0 | 1 | 0 | 1 | 0
  Week 70 | 0.7 (1.0) |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 1.0 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 71: number analyzed (Participants) | 2 | 0 | 1 | 0 | 1 | 0
  Week 71 | 0.1 (0.1) |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.8 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 72: number analyzed (Participants) | 0 | 1 | 1 | 0 | 1 | 0
  Week 72 |  | 1.2 (NA) — SD is not evaluable when only one participant is analyzed | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.9 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 73: number analyzed (Participants) | 2 | 3 | 2 | 0 | 1 | 0
  Week 73 | 0.4 (0.3) | 0.0 (0.0) | 1.3 (1.8) |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 74: number analyzed (Participants) | 3 | 0 | 1 | 0 | 1 | 0
  Week 74 | 1.3 (0.7) |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.8 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 75: number analyzed (Participants) | 2 | 0 | 1 | 0 | 1 | 0
  Week 75 | 0.2 (0.0) |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 1.1 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 76: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 76 |  |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 77: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 77 |  |  | 1.5 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.9 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 78: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0
  Week 78 | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |  | 1.4 (NA) — SD is not evaluable when only one participant is analyzed |  |  |
  Week 79: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 79 |  |  | 1.4 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.8 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 80: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0
  Week 80 | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 1.1 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.8 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 81: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Week 81 |  |  | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |  |  |
  Week 82: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Week 82 |  |  | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |  |  |
  Week 83: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 83 |  |  | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.8 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 84: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0
  Week 84 | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |  |  |
  Week 85: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 85 |  |  | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 86: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0
  Week 86 | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.6 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 89: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Week 89 |  |  |  |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0
  Week 90 | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |  |  |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Week 91 |  |  |  |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 92: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Week 92 |  |  |  |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 93: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Week 93 |  |  |  |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 94: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 94 |  |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 95: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 95 |  |  | 0.5 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 96: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 96 |  |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.8 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 97: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Week 97 |  |  |  |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 98: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 98 |  |  | 0.0 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 99: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 99 |  |  | 0.1 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 100: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 100 |  |  | 0.3 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 101: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Week 101 |  |  |  |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 102: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 102 |  |  | 0.2 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 103: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 103 |  |  | 0.3 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 104: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 104 |  |  | 0.2 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 105: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Week 105 |  |  | 0.1 (NA) — SD is not evaluable when only one participant is analyzed |  | 0.8 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 107: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Week 107 |  |  |  |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  Week 108: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Week 108 |  |  |  |  | 0.7 (NA) — SD is not evaluable when only one participant is analyzed |
  End of Treatment | 0.4 (0.6) | 0.6 (1.8) | 0.5 (0.8) | 0.8 (1.0) | 0.1 (0.2) |

ADVERSE EVENTS:
Time Frame: From Baseline up to study completion/discontinuation (up to approximately 84 months)
Description: All-Cause Mortality were reported for the ITT population. ITT population=participants who were randomized, whether or not the participants received the assigned treatment. Serious and non-serious adverse events were reported for safety population. Safety population=participants who received at least one dose of study medication.
Arm/Group | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL | Arm A (Phase II Randomization): Pola+BR in FL | Arm B (Phase II Randomization): BR in FL | Arm C (Phase II Randomization): Pola+BR in DLBCL | Arm D (Phase II Randomization): BR in DLBCL | Arm E (Phase II Expansion): Pola+BG in FL | Arm F (Phase II Expansion): Pola+BG in DLBCL | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL
All-Cause Mortality (participants affected / at risk) | 2/6 | 2/6 | 2/6 | 4/6 | 16/39 | 11/41 | 26/40 | 30/40 | 3/20 | 18/21 | 65/106
Serious Adverse Events (participants affected / at risk) | 2/6 | 4/6 | 4/6 | 5/6 | 25/38 | 12/41 | 24/39 | 27/39 | 8/20 | 13/20 | 57/106
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6 | 38/38 | 39/41 | 36/39 | 37/39 | 20/20 | 19/20 | 103/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL (N=6) | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL (N=6) | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL (N=6) | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL (N=6) | Arm A (Phase II Randomization): Pola+BR in FL (N=38) | Arm B (Phase II Randomization): BR in FL (N=41) | Arm C (Phase II Randomization): Pola+BR in DLBCL (N=39) | Arm D (Phase II Randomization): BR in DLBCL (N=39) | Arm E (Phase II Expansion): Pola+BG in FL (N=20) | Arm F (Phase II Expansion): Pola+BG in DLBCL (N=20) | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL (N=106)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (9) | 1 (1) | 4 (4) | 4 (4) | 2 (3) | 2 (2) | 9 (11)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ENTERITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 2 (3) | 7 (7)
SUDDEN DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ISCHAEMIC HEPATITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
CEREBRAL TOXOPLASMOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CYTOMEGALOVIRUS CHORIORETINITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CYTOMEGALOVIRUS ENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENTEROCOLITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GIARDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEPATITIS E (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HUMAN ANAPLASMOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFECTED LYMPHOCELE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
LARGE INTESTINE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENINGOENCEPHALITIS HERPETIC (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ORAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLEURAL INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 7 (8) | 1 (1) | 4 (4) | 4 (5) | 0 (0) | 0 (0) | 6 (6)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA CYTOMEGALOVIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA FUNGAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROGRESSIVE MULTIFOCAL LEUKOENCEPHALOPATHY (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 7 (9)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL FEVER (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EASTERN COOPERATIVE ONCOLOGY GROUP PERFORMANCE STATUS WORSENED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MORAXELLA TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LEUKOENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DISTRIBUTIVE SHOCK (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL THROMBOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENTEROCOLITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DISSEMINATED VARICELLA ZOSTER VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VASCULAR ACCESS SITE CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EPIGLOTTIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRAIN OEDEMA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in FL (N=6) | Cohort 1a (Phase Ib Safety Run-In): Pola+BR in DLBCL (N=6) | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in FL (N=6) | Cohort 1b (Phase Ib Safety Run-In): Pola+BG in DLBCL (N=6) | Arm A (Phase II Randomization): Pola+BR in FL (N=38) | Arm B (Phase II Randomization): BR in FL (N=41) | Arm C (Phase II Randomization): Pola+BR in DLBCL (N=39) | Arm D (Phase II Randomization): BR in DLBCL (N=39) | Arm E (Phase II Expansion): Pola+BG in FL (N=20) | Arm F (Phase II Expansion): Pola+BG in DLBCL (N=20) | Arm G+H (Phase II NF Cohort): Pola+BR in DLBCL (N=106)
ANAEMIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 6 (24) | 5 (5) | 10 (13) | 19 (28) | 3 (7) | 5 (6) | 27 (35)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 3 (4) | 4 (6) | 5 (19) | 0 (0) | 0 (0) | 7 (17)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 3 (4) | 0 (0) | 5 (6) | 2 (5) | 0 (0) | 5 (7)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 2 (8) | 1 (1) | 16 (31) | 11 (18) | 14 (27) | 21 (63) | 6 (10) | 6 (30) | 35 (73)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 3 (6) | 8 (13) | 11 (18) | 19 (50) | 4 (4) | 7 (10) | 19 (40)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 6 (6)
HYPOACUSIS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 5 (5) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 12 (14)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 6 (7)
APHTHOUS ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (7) | 2 (2) | 10 (10) | 8 (8) | 8 (9) | 7 (8) | 7 (11) | 9 (10) | 20 (27)
DIARRHOEA (Gastrointestinal disorders) | 2 (8) | 2 (5) | 4 (7) | 4 (4) | 16 (27) | 9 (11) | 11 (13) | 16 (28) | 10 (22) | 11 (18) | 36 (48)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 6 (6) | 2 (2) | 3 (4) | 3 (3) | 0 (0) | 5 (6)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 3 (4) | 3 (4) | 5 (7) | 3 (3) | 22 (35) | 13 (25) | 16 (19) | 12 (14) | 11 (21) | 11 (16) | 34 (38)
ODYNOPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 2 (3) | 4 (4) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (3) | 1 (2) | 5 (6) | 1 (1) | 7 (12) | 8 (11) | 5 (8) | 7 (11) | 8 (10) | 8 (10) | 17 (18)
ASTHENIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 7 (9) | 3 (5) | 6 (8) | 4 (4) | 0 (0) | 3 (3) | 12 (13)
CHILLS (General disorders) | 1 (2) | 1 (4) | 3 (5) | 2 (3) | 0 (0) | 3 (3) | 3 (4) | 4 (5) | 2 (2) | 5 (5) | 2 (2)
DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 4 (4) | 4 (5) | 3 (3) | 2 (2) | 16 (20) | 13 (22) | 14 (17) | 14 (20) | 13 (22) | 12 (15) | 22 (25)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 4 (4) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 6 (7)
PAIN (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 5 (5)
PYREXIA (General disorders) | 1 (1) | 2 (4) | 2 (4) | 2 (2) | 8 (11) | 4 (5) | 9 (15) | 10 (14) | 2 (2) | 8 (9) | 22 (27)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
HERPES VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 6 (6)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 3 (3) | 7 (7) | 1 (1) | 2 (4) | 5 (5) | 2 (3) | 7 (10)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 7 (8)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (4)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 5 (6) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 0 (0) | 4 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 5 (6)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (6) | 0 (0) | 7 (11)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (6) | 2 (2) | 4 (6) | 2 (2) | 3 (3) | 0 (0) | 4 (9)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 4 (7)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (10) | 0 (0) | 3 (5) | 1 (1) | 2 (6) | 0 (0) | 8 (16)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (15) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 14 (37)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (18) | 0 (0) | 2 (5) | 4 (5) | 1 (1) | 0 (0) | 8 (11)
WEIGHT DECREASED (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 5 (5) | 2 (3) | 1 (1) | 14 (14)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (16) | 0 (0) | 4 (6) | 1 (1) | 3 (7) | 1 (1) | 9 (29)
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 10 (13) | 5 (5) | 8 (8) | 10 (11) | 6 (7) | 8 (10) | 27 (30)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 3 (9) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 5 (7) | 1 (1) | 0 (0) | 3 (3)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 3 (5) | 2 (5) | 0 (0) | 3 (3)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (2) | 3 (3) | 2 (4) | 2 (2) | 5 (9) | 4 (6) | 3 (3) | 4 (7) | 3 (9) | 5 (5) | 15 (20)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (5) | 2 (2) | 1 (1) | 3 (3) | 4 (6) | 1 (1) | 4 (5) | 1 (1) | 4 (4) | 1 (1) | 13 (18)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (6) | 1 (1) | 1 (1) | 2 (3) | 2 (6) | 1 (1) | 2 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 3 (4) | 1 (1) | 5 (5) | 2 (4) | 1 (1) | 6 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 1 (1) | 3 (3) | 2 (2) | 7 (8)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 1 (1) | 3 (3)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 1 (2) | 3 (3) | 4 (4)
DIZZINESS (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 5 (5) | 3 (3) | 5 (5) | 3 (3) | 1 (1) | 10 (11)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 5 (5)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 8 (8) | 5 (6) | 2 (3) | 3 (3) | 6 (6) | 3 (4) | 12 (14)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (5) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (9) | 5 (5) | 1 (1) | 9 (10) | 5 (5) | 1 (1) | 15 (16)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (8) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 6 (7) | 3 (3) | 2 (2) | 5 (6)
POST HERPETIC NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 4 (4)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
INSOMNIA (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 8 (10)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (6) | 0 (0) | 6 (7) | 3 (3) | 8 (10) | 6 (6) | 2 (2) | 3 (3) | 13 (16)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (2) | 2 (3) | 4 (4) | 4 (4) | 2 (2) | 3 (3) | 7 (7) | 6 (7) | 3 (4)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 5 (6)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 2 (3)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (10)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 4 (5) | 5 (6) | 1 (1) | 0 (0) | 8 (9)
RASH (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2) | 0 (0) | 2 (2) | 3 (5) | 4 (5) | 5 (5) | 2 (2) | 3 (5) | 3 (3) | 5 (8)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 2 (2) | 1 (2) | 2 (2) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 3 (4) | 10 (12)
COAGULOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HAEMOLYSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
EYE DISCHARGE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE PRURITUS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
GLAUCOMA (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OCULAR HYPERAEMIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ANAL SPASM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEFAECATION URGENCY (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULUM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GINGIVAL DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GINGIVAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
LIP DRY (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
NONINFECTIVE GINGIVITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL DISCHARGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATHETER SITE PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATHETER SITE PRURITUS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
EARLY SATIETY (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAIT DISTURBANCE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
PERIPHERAL SWELLING (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
CANDIDA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
CYTOMEGALOVIRUS VIRAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FOLLICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 1 (1)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WOUND (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AMYLASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 4 (4)
BLOOD CALCIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD MAGNESIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
EASTERN COOPERATIVE ONCOLOGY GROUP PERFORMANCE STATUS WORSENED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
NEUTROPHIL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TROPONIN I INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TROPONIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 3 (3)
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AMNESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSKINESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERONEAL NERVE PALSY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POLYNEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SINUS HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TASTE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IRRITABILITY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
ANURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TESTICULAR PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TESTICULAR SWELLING (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
NASAL DISCHARGE DISCOLOURATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EMBOLISM (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PALLOR (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHLEBITIS SUPERFICIAL (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VASCULAR ACCESS SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT02257567/Prot_SAP_000.pdf